CLINICAL TRIAL: NCT02277106
Title: A Double-blind, Placebo-controlled, Two-Period Crossover Proof-of-Concept Study Evaluating the Safety, Tolerability, Pharmacokinetics, and Efficacy of SAGE-547 Injection in the Treatment of Patients With Essential Tremor
Brief Title: Evaluate SAGE-547 in Participants With Essential Tremor
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sage Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 547-ETD-201
Record Dates: First submitted 2014-10-22; First posted 2014-10-28 (Estimated); Results first posted 2022-06-29 (Actual); Last update posted 2022-06-29 (Actual); Status verified 2022-06

CONDITIONS: Essential Tremor
MeSH Terms: conditions — Essential Tremor | interventions — brexanolone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Stage 1 (Double-blind): SAGE 547, Then Placebo (Experimental): Participants received a 12-hour intravenous (IV) infusion of SAGE 547, at ascending doses of 29, 58, and 86 micrograms per kilogram of body weight per hour (μg/kg/h), 4 hours each, on Day 1 of Stage 1 [Treatment Period 1 (TP 1)]. After a washout period of approximately 7 days, participants received a 12-hour IV infusion of SAGE-547 matching-placebo, on Day 10 of Stage 1 [Treatment Period 2 (TP 2)].
  Interventions: Drug: SAGE-547; Drug: Placebo
- Stage 1 (Double-blind): Placebo, Then SAGE-547 (Experimental): Participants received a 12-hour IV infusion of SAGE-547 matching-placebo on Day 1 of Stage 1 (TP 1). After a washout period of approximately 7 days, participants received a 12-hour IV infusion of SAGE 547 at ascending doses of 29, 58, and 86 μg/kg/h, 4 hours each, on Day 10 of Stage 1 (TP 2).
  Interventions: Drug: SAGE-547; Drug: Placebo
- Stage 2 (Open Label): SAGE-547 (Experimental): Participants who completed Stage 1 were invited to receive a 10-hour IV infusion of SAGE 547, at ascending doses of 90 μg/kg/h for 1 hour, 120 μg/kg/h for 1 hour, and 150 μg/kg/h for 8 hours on Day 1 of Stage 2.
  Interventions: Drug: SAGE-547

INTERVENTIONS:
Drug: SAGE-547
Drug: Placebo
  Arms: Stage 1 (Double-blind): Placebo, Then SAGE-547; Stage 1 (Double-blind): SAGE 547, Then Placebo

SUMMARY:
Stage 1 is a double-blind, proof-of-concept study designed to evaluate the safety, tolerability, pharmacokinetics (PK), and efficacy of SAGE-547 Injection in male and female participants with essential tremor in the upper limb.

Stage 2 is an open-label arm designed to evaluate the safety, tolerability, PK, and effectiveness of SAGE-547 Injection at a higher dose than in Stage 1. Participants who completed Stage 1 were invited to participate in Stage 2.

ELIGIBILITY:
Inclusion Criteria:

* Males and females, 35-75 years old with a diagnosis of essential tremor with symptoms clearly present in at least 1 upper limb; participant has had tremor present for at least 2 years prior to Screening
* Off medication, or on a stable dose of medication for their tremor for at least 28 days prior to Screening

Exclusion Criteria:

* Recent history or active clinically significant manifestations of metabolic, hepatic, renal, hematological, pulmonary, cardiovascular, gastrointestinal, musculoskeletal, dermatological, urogenital, eyes, ears, nose, or throat, psychiatric, or neurological (other than essential tremor) disorders
* Medical history of seizures

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2014-09-23 (Actual); Primary Completion 2015-08-14 (Actual); Study Completion 2015-08-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Lasser, MD, MBA, Study Chair — Sage Therapeutics
Locations (2):
- United States (2):
  - Sage Study Site, Bingham Farms, Michigan
  - Sage Study Site, Raleigh, North Carolina

IPD SHARING:
Plan to Share IPD: No
Data sharing will be consistent with the results submission policy of ClinicalTrials.gov.

REFERENCES:
- [Result] Aaron Ellenbogen, Shane Raines, Stephen Kanes. Exploratory trial results for SAGE-547 in essential tremor. Presented at AAN, April 19, 2016 P4.297. MRC-ZUL-00141_Exploratory Trial Results for SAGE-547 in Essential Tremor.
- See also: Sage Therapeutics — http://www.sagerx.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 2 investigative sites in the United States from 23 September 2014 to 14 August 2015.
Pre-assignment Details: This study consisted of two stages, Stages 1 and 2. Stage 1 had two periods with treatment on Days 1 and 10 and a 7-day follow-up period. Participants were followed for serious adverse events (SAEs) up to 30 days after the last dose. Stage 2 follows Stage 1, with treatment on Day 1 and a 7-day follow-up period thereafter.
Period: Stage 1: Treatment Period 1
Arm/Group | Stage 1 (Double-blind): SAGE 547, Then Placebo | Stage 1 (Double-blind): Placebo, Then SAGE-547 | Stage 2 (Open Label): SAGE-547
Started | 13 | 12 | 0
Completed | 13 | 12 | 0
Not Completed | 0 | 0 | 0
Period: Washout
Arm/Group | Stage 1 (Double-blind): SAGE 547, Then Placebo | Stage 1 (Double-blind): Placebo, Then SAGE-547 | Stage 2 (Open Label): SAGE-547
Started | 13 | 12 | 0
Completed | 13 | 12 | 0
Not Completed | 0 | 0 | 0
Period: Stage 1: Treatment Period 2
Arm/Group | Stage 1 (Double-blind): SAGE 547, Then Placebo | Stage 1 (Double-blind): Placebo, Then SAGE-547 | Stage 2 (Open Label): SAGE-547
Started | 13 | 12 | 0
Completed | 13 | 12 | 0
Not Completed | 0 | 0 | 0
Period: Stage 2
Arm/Group | Stage 1 (Double-blind): SAGE 547, Then Placebo | Stage 1 (Double-blind): Placebo, Then SAGE-547 | Stage 2 (Open Label): SAGE-547
Started | 0 | 0 | 17 (Out of 25, 17 participants entered Stage 2 after Screening at Stage 2.)
Completed | 0 | 0 | 16
Not Completed | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety population included all participants admitted into the inpatient unit who met all eligibility criteria, signed an informed consent, and who began infusion with SAGE-547 or placebo in Treatment Period 1 of Stage 1.
Groups:
- Stage 1 (Double-blind): SAGE-547 and Placebo: Participants who received a 12-hour IV infusion of SAGE 547, at ascending doses of 29, 58, and 86 μg/kg/h, 4 hours each, on Day 1 of Stage 1 (TP 1), received a 12-hour IV infusion of SAGE-547 matched-placebo, on Day 10 of Stage 1 (TP 2), after a washout period of approximately 7 days. Participants who received a 12-hour IV infusion of SAGE-547 matched-placebo on Day 1 of Stage 1 (TP 1), received a 12-hour IV infusion of SAGE 547 at ascending doses of 29, 58, and 86 μg/kg/h, 4 hours each, on Day 10 of Stage 1 (TP 2), after a washout period of approximately 7 days.
Arm/Group | Stage 1 (Double-blind): SAGE-547 and Placebo
Number analyzed (Participants) | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.2 (5.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 24
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 1
  White | 22
  Other | 2

OUTCOME MEASURES:

1. Primary Outcome: Stage 1: Percentage of Participants With Treatment-Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Description: An adverse event (AE) is any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug related. A TEAE was defined as an AE with start date/time after the start of initial infusion in each stage. An SAE is defined as an AE or suspected adverse reaction, which in the view of either the Investigator or Sponsor, results in any of the following outcomes: death; is life-threatening; inpatient hospitalization or prolongation of existing hospitalization; a persistent or significant disability or incapacity; congenital anomaly or birth defect or other medically important condition.
Time Frame: Stage 1: Up to 30 days after last infusion (up to Day 40)
Population: as for baseline characteristics
Measure: Number; unit: percentage of participants
Groups:
- Stage 1: SAGE-547: Participants received a 12-hour IV infusion of SAGE 547, at ascending doses of 29, 58, and 86 μg/kg/h, 4 hours each, on Day 1 of Stage 1 (TP 1) or on Day 10 of Stage 1 (TP 2).
- Stage 1: Placebo: Participants received a 12-hour IV infusion of SAGE-547 matching-placebo on Day 1 of Stage 1 (TP 1) or on Day 10 of Stage 1 (TP 2).
Arm/Group | Stage 1: SAGE-547 | Stage 1: Placebo
Number analyzed (Participants) | 25 | 25
percentage of participants
  TEAEs | 12.0 | 20.0
  SAEs | 0 | 0

2. Primary Outcome: Stage 2: Percentage of Participants With Treatment-Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Description: An AE is any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug related. A TEAE was defined as an AE with start date/time after the start of initial infusion in each stage. An SAE is defined as an AE or suspected adverse reaction, which in the view of either the Investigator or Sponsor, results in any of the following outcomes: death; is life-threatening; inpatient hospitalization or prolongation of existing hospitalization; a persistent or significant disability or incapacity; congenital anomaly or birth defect or other medically important condition.
Time Frame: Stage 2: Up to 30 days after last infusion (up to Day 31)
Population: Participants from safety population, which included all participants admitted into the inpatient unit who met all eligibility criteria, signed an informed consent, and who began infusion with SAGE-547 or placebo in Treatment Period 1, who received study drug in Stage 2.
Measure: Number; unit: percentage of participants
Groups:
- Stage 2: SAGE-547: Participants who completed Stage 1 received a 10-hour IV infusion of SAGE 547, at ascending doses of 90 μg/kg/h for 1 hour, 120 μg/kg/h for 1 hour, and 150 μg/kg/h for 8 hours on Day 1 of Stage 2.
Arm/Group | Stage 2: SAGE-547
Number analyzed (Participants) | 17
percentage of participants
  TEAEs | 47.1
  SAEs | 0

3. Primary Outcome: Stage 1: Percentage of Participants With a Response of 'Yes' to Any Columbia Suicide Severity Rating Scale (C-SSRS) Suicidal Ideation or Suicidal Behavior Item at Any Visit
Description: The C-SSRS scale consisted of baseline evaluation that assessed lifetime experience of participants with suicidal ideation (SI) and suicidal behavior (SB) and postbaseline evaluation that focused on suicidality since last study visit. C-SSRS included "yes" or "no"' responses for assessment of suicidal ideation and behavior as well as numeric ratings for severity of ideation, if present [from 1 (minor physical damage) to 5 (death), with 5 being most severe]. C-SSRS SI items involved (a) wish to be dead, (b) non-specific active suicidal thoughts, (c) active SI with any methods (not plan) without intent to act, (d) active SI with some intent to act, without specific plan and (e) active SI with specific plan and intent. C-SSRS SB items involved (a) actual attempt, (b) engaged in non-suicidal self-injurious behavior, (c) interrupted attempt, (d) aborted attempt, (e) preparatory acts or behavior, (f) suicidal behavior. Only categories with data are reported.
Time Frame: Stage 1: Pre-infusion on Day 1 of Stage 1 (Treatment Period 1) or on Day 10 of Stage 1 (Treatment Period 2)
Population: as for baseline characteristics
Measure: Number; unit: percentage of participants
Groups:
- Stage 1: Placebo: Participants received one 12-hour IV infusion of SAGE-547 matching-placebo on Day 1 of Stage 1 (TP 1) or on Day 10 of Stage 1 (TP 2).
Arm/Group | Stage 1: SAGE-547 | Stage 1: Placebo
Number analyzed (Participants) | 25 | 25
percentage of participants
  Suicidal Ideation: Wish to be Dead: Pre-infusion | 0 | 4.0
  Suicidal Ideation: Non-specific Active Suicidal Thoughts: Pre-infusion | 4.0 | 0
  Suicidal Behavior: Actual Attempt: Pre-infusion | 4.0 | 4.0

4. Primary Outcome: Stage 2: Percentage of Participants With a Response of 'Yes' to Any Columbia Suicide Severity Rating Scale (C-SSRS) Suicidal Ideation or Suicidal Behavior Item at Any Visit
Description: The C-SSRS scale consisted of baseline evaluation that assessed lifetime experience of participants with SI and SB and postbaseline evaluation that focused on suicidality since last study visit. C-SSRS included "yes" or "no"' responses for assessment of suicidal ideation and behavior as well as numeric ratings for severity of ideation, if present [from 1 (minor physical damage) to 5 (death), with 5 being most severe]. C-SSRS SI items involved (a) wish to be dead, (b) non-specific active suicidal thoughts, (c) active SI with any methods (not plan) without intent to act, (d) active SI with some intent to act, without specific plan and (e) active SI with specific plan and intent. C-SSRS SB items involved (a) actual attempt, (b) engaged in non-suicidal self-injurious behavior, (c) interrupted attempt, (d) aborted attempt, (e) preparatory acts or behavior, (f) suicidal behavior.
Time Frame: Stage 2 Day 1: Pre-infusion and 10 hours and 7-day follow-up post-infusion
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Groups:
- Stage 2: SAGE-547: Participants who completed Stage 1 were invited to receive a 10-hour IV infusion of SAGE 547, at ascending doses of 90 μg/kg/h for 1 hour, 120 μg/kg/h for 1 hour, and 150 μg/kg/h for 8 hours on Day 1 of Stage 2.
Arm/Group | Stage 2: SAGE-547
Number analyzed (Participants) | 17
percentage of participants | 0

5. Primary Outcome: Stage 1: Change From Baseline (CFB) in Vital Signs Parameter - Supine Systolic Blood Pressure
Description: Vital signs included supine systolic blood pressure, supine diastolic blood pressure, supine heart rate, standing systolic blood pressure, standing diastolic blood pressure, standing heart rate, temperature, and respiratory rate. CFB in supine systolic blood pressure is reported in this outcome measure. Baseline is defined as the pre-infusion value in each period/stage.
Time Frame: Day 1 of Stage 1 (Treatment Period 1) or on Day 10 of Stage 1 (Treatment Period 2): Pre-infusion (Baseline) and 4, 8, 12 hours during infusion and 12-hour follow-up post-infusion
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: millimeters of mercury (mmHg)
Arm/Group | Stage 1: SAGE-547 | Stage 1: Placebo
Number analyzed (Participants) | 25 | 25
millimeters of mercury (mmHg)
  Pre-infusion | 121.6 (11.58) | 120.2 (15.47)
  CFB at 4 Hours | -2.5 (10.84) | 4.0 (11.71)
  CFB at 8 Hours | -3.9 (11.64) | 3.5 (10.24)
  CFB at 12 Hours | -1.6 (10.44) | 7.6 (10.14)
  CFB at 12-hour Follow-up | 5.6 (8.68) | 1.4 (11.85)

6. Primary Outcome: Stage 2: Change From Baseline in Vital Signs Parameter - Supine Systolic Blood Pressure
Description: as for outcome 5
Time Frame: Stage 2 Day 1: Pre-infusion (Baseline) and 2, 4, 6, 8, 10, 12, 14 and 24 hours post-infusion
Population: Participants from safety population, which included all participants admitted into the inpatient unit who met all eligibility criteria, signed an informed consent, and who began infusion with SAGE-547 or placebo in Treatment Period 1, who received study drug in Stage 2. Number analyzed = Number of participants with data available at the specific time point.
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- Stage 2: SAGE-547: Participants who completed Stage 1 received one 10-hour IV infusion of SAGE 547, at ascending doses of 90 μg/kg/h for 1 hour, 120 μg/kg/h for 1 hour, and 150 μg/kg/h for 8 hours on Day 1 of Stage 2.
Arm/Group | Stage 2: SAGE-547
Number analyzed (Participants) | 17
mmHg
  Pre-infusion | 125.3 (13.22)
  CFB at 2 Hours | -12.1 (14.95)
  CFB at 4 Hours: number analyzed (Participants) | 16
  CFB at 4 Hours | -7.6 (17.12)
  CFB at 6 Hours: number analyzed (Participants) | 16
  CFB at 6 Hours | -7.9 (14.01)
  CFB at 8 Hours: number analyzed (Participants) | 16
  CFB at 8 Hours | -6.8 (17.44)
  CFB at 10 Hours: number analyzed (Participants) | 16
  CFB at 10 Hours | -2.9 (13.48)
  CFB at 12 Hours: number analyzed (Participants) | 16
  CFB at 12 Hours | 4.0 (13.22)
  CFB at 14 Hours: number analyzed (Participants) | 16
  CFB at 14 Hours | 3.1 (18.44)
  CFB at 24 Hours: number analyzed (Participants) | 16
  CFB at 24 Hours | 4.3 (11.12)

7. Primary Outcome: Stage 1: Change From Baseline in Vital Signs Parameter - Supine Diastolic Blood Pressure
Description: Vital signs included supine systolic blood pressure, supine diastolic blood pressure, supine heart rate, standing systolic blood pressure, standing diastolic blood pressure, standing heart rate, temperature, and respiratory rate. CFB in supine diastolic blood pressure is reported in this outcome measure. Baseline is defined as the pre-infusion value in each period/stage.
Time Frame: as for outcome 5
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Stage 1: SAGE-547 | Stage 1: Placebo
Number analyzed (Participants) | 25 | 25
mmHg
  Pre-infusion | 74.3 (8.90) | 75.0 (11.24)
  CFB at 4 Hours | -2.3 (9.85) | -0.6 (6.10)
  CFB at 8 Hours | -2.0 (6.79) | -0.7 (8.27)
  CFB at 12 Hours | 0.4 (8.33) | 1.2 (9.69)
  CFB at 12-hour Follow-up | 2.0 (8.17) | 0.8 (9.68)

8. Primary Outcome: Stage 2: Change From Baseline in Vital Signs Parameter - Supine Diastolic Blood Pressure
Description: as for outcome 7
Time Frame: Stage 2 Day 1: Pre-infusion (Baseline) and 2, 4, 6, 8, 10, 12, 14 and 24 hours post-infusion
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Stage 2: SAGE-547
Number analyzed (Participants) | 17
mmHg
  Pre-infusion | 75.5 (7.63)
  CFB at 2 Hours | -7.9 (8.59)
  CFB at 4 Hours: number analyzed (Participants) | 16
  CFB at 4 Hours | -6.4 (10.20)
  CFB at 6 Hours: number analyzed (Participants) | 16
  CFB at 6 Hours | -4.6 (9.70)
  CFB at 8 Hours: number analyzed (Participants) | 16
  CFB at 8 Hours | -8.8 (10.17)
  CFB at 10 Hours: number analyzed (Participants) | 16
  CFB at 10 Hours | -2.4 (9.52)
  CFB at 12 Hours: number analyzed (Participants) | 16
  CFB at 12 Hours | 0.3 (8.80)
  CFB at 14 Hours: number analyzed (Participants) | 16
  CFB at 14 Hours | -2.2 (9.03)
  CFB at 24 Hours: number analyzed (Participants) | 16
  CFB at 24 Hours | -0.3 (8.99)

9. Primary Outcome: Stage 1: Change From Baseline in Vital Signs Parameter - Supine Heart Rate
Description: Vital signs included supine systolic blood pressure, supine diastolic blood pressure, supine heart rate, standing systolic blood pressure, standing diastolic blood pressure, standing heart rate, temperature, and respiratory rate. CFB in supine heart rate is reported in this outcome measure. Baseline is defined as the pre-infusion value in each period/stage.
Time Frame: as for outcome 5
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: beats per minute (bpm)
Arm/Group | Stage 1: SAGE-547 | Stage 1: Placebo
Number analyzed (Participants) | 25 | 25
beats per minute (bpm)
  Pre-infusion | 66.0 (9.70) | 69.0 (12.99)
  CFB at 4 Hours | -1.4 (7.52) | -2.1 (10.39)
  CFB at 8 Hours | 2.0 (6.37) | 1.3 (14.85)
  CFB at 12 Hours | 5.0 (8.67) | 2.1 (11.23)
  CFB at 12-hour Follow-up | 2.9 (9.17) | -2.3 (8.96)

10. Primary Outcome: Stage 2: Change From Baseline in Vital Signs Parameter - Supine Heart Rate
Description: as for outcome 9
Time Frame: Stage 2 Day 1: Pre-infusion (Baseline) and 2, 4, 6, 8, 10, 12, 14 and 24 hours post-infusion
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | Stage 2: SAGE-547
Number analyzed (Participants) | 17
bpm
  Pre-infusion | 69.5 (10.96)
  CFB at 2 Hours | 0.7 (10.18)
  CFB at 4 Hours: number analyzed (Participants) | 16
  CFB at 4 Hours | -3.3 (7.22)
  CFB at 6 Hours: number analyzed (Participants) | 16
  CFB at 6 Hours | -3.3 (10.30)
  CFB at 8 Hours: number analyzed (Participants) | 16
  CFB at 8 Hours | -1.5 (9.00)
  CFB at 10 Hours: number analyzed (Participants) | 16
  CFB at 10 Hours | -1.5 (9.10)
  CFB at 12 Hours: number analyzed (Participants) | 16
  CFB at 12 Hours | -2.1 (8.55)
  CFB at 14 Hours: number analyzed (Participants) | 16
  CFB at 14 Hours | 3.9 (10.29)
  CFB at 24 Hours: number analyzed (Participants) | 16
  CFB at 24 Hours | 2.6 (8.70)

11. Primary Outcome: Stage 1: Change From Baseline in Vital Signs Parameter - Standing Systolic Blood Pressure
Description: Vital signs included supine systolic blood pressure, supine diastolic blood pressure, supine heart rate, standing systolic blood pressure, standing diastolic blood pressure, standing heart rate, temperature, and respiratory rate. CFB in standing systolic blood pressure is reported in this outcome measure. Baseline is defined as the pre-infusion value in each period/stage.
Time Frame: as for outcome 5
Population: Safety population included all participants admitted into the inpatient unit who met all eligibility criteria, signed an informed consent, and who began infusion with SAGE-547 or placebo in Treatment Period 1 of Stage 1 .
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Stage 1: SAGE-547 | Stage 1: Placebo
Number analyzed (Participants) | 25 | 25
mmHg
  Pre-infusion | 118.0 (17.27) | 119.1 (15.00)
  CFB at 4 Hours | -2.2 (10.70) | 1.7 (12.48)
  CFB at 8 Hours | -2.7 (13.23) | 1.0 (12.87)
  CFB at 12 Hours | 2.0 (12.65) | 7.8 (11.48)
  CFB at 12-hour Follow-up | 5.0 (15.82) | 1.7 (10.76)

12. Primary Outcome: Stage 2: Change From Baseline in Vital Signs Parameter - Standing Systolic Blood Pressure
Description: as for outcome 11
Time Frame: Stage 2 Day 1: Pre-infusion (Baseline) and 2, 4, 6, 8, 10, 12, 14 and 24 hours post-infusion
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Stage 2: SAGE-547
Number analyzed (Participants) | 17
mmHg
  Pre-infusion | 120.1 (13.05)
  CFB at 2 Hours | -5.5 (15.98)
  CFB at 4 Hours: number analyzed (Participants) | 16
  CFB at 4 Hours | -5.9 (13.87)
  CFB at 6 Hours: number analyzed (Participants) | 16
  CFB at 6 Hours | -1.0 (16.84)
  CFB at 8 Hours: number analyzed (Participants) | 16
  CFB at 8 Hours | -2.9 (14.22)
  CFB at 10 Hours: number analyzed (Participants) | 16
  CFB at 10 Hours | -0.9 (16.49)
  CFB at 12 Hours: number analyzed (Participants) | 16
  CFB at 12 Hours | 10.2 (17.28)
  CFB at 14 Hours: number analyzed (Participants) | 16
  CFB at 14 Hours | 11.1 (18.98)
  CFB at 24 Hours: number analyzed (Participants) | 16
  CFB at 24 Hours | 2.9 (9.30)

13. Primary Outcome: Stage 1: Change From Baseline in Vital Signs Parameter - Standing Diastolic Blood Pressure
Description: Vital signs included supine systolic blood pressure, supine diastolic blood pressure, supine heart rate, standing systolic blood pressure, standing diastolic blood pressure, standing heart rate, temperature, and respiratory rate. CFB in standing diastolic blood pressure is reported in this outcome measure. Baseline is defined as the pre-infusion value in each period/stage.
Time Frame: as for outcome 5
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Stage 1: SAGE-547 | Stage 1: Placebo
Number analyzed (Participants) | 25 | 25
mmHg
  Pre-infusion | 76.2 (10.20) | 78.9 (11.84)
  CFB at 4 Hours | -1.2 (8.86) | -3.1 (6.81)
  CFB at 8 Hours | -2.1 (9.03) | -2.6 (7.34)
  CFB at 12 Hours | 1.0 (9.53) | 0.6 (9.31)
  CFB at 12-hour Follow-up | 2.7 (9.85) | 0.9 (6.65)

14. Primary Outcome: Stage 2: Change From Baseline in Vital Signs Parameter - Standing Diastolic Blood Pressure
Description: as for outcome 13
Time Frame: Stage 2 Day 1: Pre-infusion (Baseline) and 2, 4, 6, 8, 10, 12, 14 and 24 hours post-infusion
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Stage 2: SAGE-547
Number analyzed (Participants) | 17
mmHg
  Pre-infusion | 78.9 (8.81)
  CFB at 2 Hours | -5.6 (7.17)
  CFB at 4 Hours: number analyzed (Participants) | 16
  CFB at 4 Hours | -4.5 (8.43)
  CFB at 6 Hours: number analyzed (Participants) | 16
  CFB at 6 Hours | -4.1 (6.66)
  CFB at 8 Hours: number analyzed (Participants) | 16
  CFB at 8 Hours | -4.7 (6.03)
  CFB at 10 Hours: number analyzed (Participants) | 16
  CFB at 10 Hours | -4.3 (9.21)
  CFB at 12 Hours: number analyzed (Participants) | 16
  CFB at 12 Hours | -1.3 (8.30)
  CFB at 14 Hours: number analyzed (Participants) | 16
  CFB at 14 Hours | -0.6 (8.73)
  CFB at 24 Hours: number analyzed (Participants) | 16
  CFB at 24 Hours | -1.5 (6.52)

15. Primary Outcome: Stage 1: Change From Baseline in Vital Signs Parameter - Standing Heart Rate
Description: Vital signs included supine systolic blood pressure, supine diastolic blood pressure, supine heart rate, standing systolic blood pressure, standing diastolic blood pressure, standing heart rate, temperature, and respiratory rate. CFB in standing heart rate is reported in this outcome measure. Baseline is defined as the pre-infusion value in each period/stage.
Time Frame: as for outcome 5
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | Stage 1: SAGE-547 | Stage 1: Placebo
Number analyzed (Participants) | 25 | 25
bpm
  Pre-infusion | 72.0 (9.66) | 75.6 (13.70)
  CFB at 4 Hours | 0.0 (7.13) | -1.0 (9.17)
  CFB at 8 Hours | 3.0 (7.55) | -0.0 (10.22)
  CFB at 12 Hours | 5.4 (11.84) | 3.4 (8.23)
  CFB at 12-hour Follow-up | 3.8 (8.15) | -1.5 (9.38)

16. Primary Outcome: Stage 2: Change From Baseline in Vital Signs Parameter - Standing Heart Rate
Description: as for outcome 15
Time Frame: Stage 2 Day 1: Pre-infusion (Baseline) and 2, 4, 6, 8, 10, 12, 14 and 24 hours post-infusion
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | Stage 2: SAGE-547
Number analyzed (Participants) | 17
bpm
  Pre-infusion | 74.6 (10.12)
  CFB at 2 Hours | 1.2 (9.25)
  CFB at 4 Hours: number analyzed (Participants) | 16
  CFB at 4 Hours | 0.7 (7.69)
  CFB at 6 Hours: number analyzed (Participants) | 16
  CFB at 6 Hours | -1.2 (7.06)
  CFB at 8 Hours: number analyzed (Participants) | 16
  CFB at 8 Hours | 2.6 (11.09)
  CFB at 10 Hours: number analyzed (Participants) | 16
  CFB at 10 Hours | 3.5 (8.53)
  CFB at 12 Hours: number analyzed (Participants) | 16
  CFB at 12 Hours | -1.5 (6.26)
  CFB at 14 Hours: number analyzed (Participants) | 16
  CFB at 14 Hours | 2.3 (10.02)
  CFB at 24 Hours: number analyzed (Participants) | 16
  CFB at 24 Hours | 4.6 (11.17)

17. Primary Outcome: Stage 1: Change From Baseline in Vital Signs Parameter - Temperature
Description: Vital signs included supine systolic blood pressure, supine diastolic blood pressure, supine heart rate, standing systolic blood pressure, standing diastolic blood pressure, standing heart rate, temperature, and respiratory rate. CFB in temperature is reported in this outcome measure. Baseline is defined as the pre-infusion value in each period/stage.
Time Frame: as for outcome 5
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: degree Celsius
Arm/Group | Stage 1: SAGE-547 | Stage 1: Placebo
Number analyzed (Participants) | 25 | 25
degree Celsius
  Pre-infusion | 36.62 (0.14) | 36.58 (0.16)
  CFB at 4 Hours | -0.03 (0.22) | 0.05 (0.25)
  CFB at 8 Hours | -0.04 (0.16) | 0.06 (0.28)
  CFB at 12 Hours | -0.02 (0.20) | 0.04 (0.23)
  CFB at 12-hour Follow-up | -0.01 (0.22) | -0.00 (0.23)

18. Primary Outcome: Stage 2: Change From Baseline in Vital Signs Parameter - Temperature
Description: as for outcome 17
Time Frame: Stage 2 Day 1: Pre-infusion (Baseline) and 2, 4, 6, 8, 10, 12, 14 and 24 hours post-infusion
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: degree Celsius
Arm/Group | Stage 2: SAGE-547
Number analyzed (Participants) | 17
degree Celsius
  Pre-infusion | 36.64 (0.15)
  CFB at 2 Hours | -0.01 (0.25)
  CFB at 4 Hours: number analyzed (Participants) | 16
  CFB at 4 Hours | -0.06 (0.20)
  CFB at 6 Hours: number analyzed (Participants) | 16
  CFB at 6 Hours | 0.01 (0.18)
  CFB at 8 Hours: number analyzed (Participants) | 16
  CFB at 8 Hours | -0.02 (0.23)
  CFB at 10 Hours: number analyzed (Participants) | 16
  CFB at 10 Hours | 0.02 (0.20)
  CFB at 12 Hours: number analyzed (Participants) | 16
  CFB at 12 Hours | -0.01 (0.40)
  CFB at 14 Hours: number analyzed (Participants) | 16
  CFB at 14 Hours | 0.02 (0.21)
  CFB at 24 Hours: number analyzed (Participants) | 16
  CFB at 24 Hours | -0.01 (0.29)

19. Primary Outcome: Stage 1: Change From Baseline in Vital Signs Parameter - Respiratory Rate
Description: Vital signs included supine systolic blood pressure, supine diastolic blood pressure, supine heart rate, standing systolic blood pressure, standing diastolic blood pressure, standing heart rate, temperature, and respiratory rate. CFB in respiratory rate is reported in this outcome measure. Baseline is defined as the pre-infusion value in each period/stage.
Time Frame: as for outcome 5
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: breaths per minute (breaths/min)
Arm/Group | Stage 1: SAGE-547 | Stage 1: Placebo
Number analyzed (Participants) | 25 | 25
breaths per minute (breaths/min)
  Pre-infusion | 16.0 (1.53) | 16.3 (1.46)
  CFB at 4 Hours | 0.4 (2.55) | -0.2 (1.52)
  CFB at 8 Hours | 0.7 (2.43) | 0.3 (2.30)
  CFB at 12 Hours | 1.0 (2.30) | 0.4 (2.04)
  CFB at 12-hour Follow-up | 0.4 (1.70) | 0.2 (1.31)

20. Primary Outcome: Stage 2: Change From Baseline in Vital Signs Parameter - Respiratory Rate
Description: as for outcome 19
Time Frame: Stage 2 Day 1: Pre-infusion (Baseline) and 2, 4, 6, 8, 10, 12, 14 and 24 hours post-infusion
Population: Participants from safety population, which included all participants admitted into the inpatient unit who met all eligibility criteria, signed an informed consent, and who began infusion with SAGE-547 or placebo in Treatment Period 1, who received study drug in Stage 2. Overall number of participants analyzed = Number of participants analyzed in this outcome measure. Number analyzed = Number of participants with data available at the specific time point.
Measure: Mean (Standard Deviation); unit: breaths/min
Arm/Group | Stage 2: SAGE-547
Number analyzed (Participants) | 17
breaths/min
  Pre-infusion | 16.9 (1.75)
  CFB at 2 Hours | -0.5 (1.81)
  CFB at 4 Hours: number analyzed (Participants) | 16
  CFB at 4 Hours | -0.4 (2.22)
  CFB at 6 Hours: number analyzed (Participants) | 16
  CFB at 6 Hours | -0.9 (2.31)
  CFB at 8 Hours: number analyzed (Participants) | 16
  CFB at 8 Hours | -0.4 (1.82)
  CFB at 10 Hours: number analyzed (Participants) | 16
  CFB at 10 Hours | 0.3 (1.24)
  CFB at 12 Hours: number analyzed (Participants) | 16
  CFB at 12 Hours | 0.5 (2.13)
  CFB at 14 Hours: number analyzed (Participants) | 16
  CFB at 14 Hours | 0.1 (2.33)
  CFB at 24 Hours: number analyzed (Participants) | 16
  CFB at 24 Hours | -0.5 (2.00)

21. Primary Outcome: Stage 1: Change From Baseline in Serum Chemistry Parameter - Alanine Aminotransferase Levels
Description: Serum chemistry parameters included alanine aminotransferase, aspartate aminotransferase, gamma glutamyl transferase, sodium, potassium, calcium, chloride, bicarbonate, protein, glucose, lactate dehydrogenase, cholesterol, triglycerides, albumin, bilirubin, creatinine, blood urea nitrogen, alkaline phosphatase, creatinine kinase, phosphate, and urate. CFB in alanine aminotransferase levels is reported in this outcome measure. Baseline is defined as the pre-infusion value in each period/stage.
Time Frame: Day 1 of Stage 1 (Treatment Period 1) or on Day 10 of Stage 1 (Treatment Period 2): Pre-infusion (Baseline) and 12-hour follow-up post-infusion
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: units per liter (u/L)
Arm/Group | Stage 1: SAGE-547 | Stage 1: Placebo
Number analyzed (Participants) | 25 | 25
units per liter (u/L)
  Pre-infusion | 22.0 (12.15) | 23.3 (14.67)
  CFB at 12-hour Follow-up | -1.4 (4.05) | -2.7 (5.69)

22. Primary Outcome: Stage 2: Absolute Values of Serum Chemistry Parameter - Alanine Aminotransferase Levels
Description: Serum chemistry parameters included alanine aminotransferase, aspartate aminotransferase, gamma glutamyl transferase, sodium, potassium, calcium, chloride, bicarbonate, protein, glucose, lactate dehydrogenase, cholesterol, triglycerides, albumin, bilirubin, creatinine, blood urea nitrogen, alkaline phosphatase, creatinine kinase, phosphate, and urate. Absolute values for alanine aminotransferase levels are reported in this outcome measure.
Time Frame: Stage 2: Any day in Screening period (Day -7 up to Day -1) and any day in 7-day follow up
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: u/L
Arm/Group | Stage 2: SAGE-547
Number analyzed (Participants) | 17
u/L
  Any Day in Screening Period (Day -7 up to Day -1) | 23.1 (11.81)
  Any Day in 7-day Follow-up | 23.6 (13.06)

23. Primary Outcome: Stage 1: Change From Baseline in Serum Chemistry Parameter - Aspartate Aminotransferase Levels
Description: Serum chemistry parameters included alanine aminotransferase, aspartate aminotransferase, gamma glutamyl transferase, sodium, potassium, calcium, chloride, bicarbonate, protein, glucose, lactate dehydrogenase, cholesterol, triglycerides, albumin, bilirubin, creatinine, blood urea nitrogen, alkaline phosphatase, creatinine kinase, phosphate, and urate. CFB in aspartate aminotransferase levels is reported in this outcome measure. Baseline is defined as the pre-infusion value in each period/stage.
Time Frame: as for outcome 21
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: u/L
Arm/Group | Stage 1: SAGE-547 | Stage 1: Placebo
Number analyzed (Participants) | 25 | 25
u/L
  Pre-infusion | 19.2 (6.31) | 19.0 (5.81)
  CFB at 12-hour Follow-up | -0.7 (3.92) | -0.0 (4.32)

24. Primary Outcome: Stage 2: Absolute Values of Serum Chemistry Parameter - Aspartate Aminotransferase Levels
Description: Serum chemistry parameters included alanine aminotransferase, aspartate aminotransferase, gamma glutamyl transferase, sodium, potassium, calcium, chloride, bicarbonate, protein, glucose, lactate dehydrogenase, cholesterol, triglycerides, albumin, bilirubin, creatinine, blood urea nitrogen, alkaline phosphatase, creatinine kinase, phosphate, and urate. Absolute values for aspartate aminotransferase levels are reported in this outcome measure.
Time Frame: Stage 2: Any day in Screening period (Day -7 up to Day -1) and any day in 7-day follow up
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: u/L
Arm/Group | Stage 2: SAGE-547
Number analyzed (Participants) | 17
u/L
  Any Day in Screening Period (Day -7 up to Day -1) | 15.8 (4.82)
  Any Day in 7-day Follow-up | 15.6 (5.66)

25. Primary Outcome: Stage 1: Change From Baseline in Serum Chemistry Parameter - Gamma Glutamyl Transferase Levels
Description: Serum chemistry parameters included alanine aminotransferase, aspartate aminotransferase, gamma glutamyl transferase, sodium, potassium, calcium, chloride, bicarbonate, protein, glucose, lactate dehydrogenase, cholesterol, triglycerides, albumin, bilirubin, creatinine, blood urea nitrogen, alkaline phosphatase, creatinine kinase, phosphate, and urate. CFB in gamma glutamyl transferase levels is reported in this outcome measure. Baseline is defined as the pre-infusion value in each period/stage.
Time Frame: as for outcome 21
Population: Safety population included all participants admitted into the inpatient unit who met all eligibility criteria, signed an informed consent, and who began infusion with SAGE-547 or placebo in Treatment Period 1 Stage 1.
Measure: Mean (Standard Deviation); unit: u/L
Arm/Group | Stage 1: SAGE-547 | Stage 1: Placebo
Number analyzed (Participants) | 25 | 25
u/L
  Pre-infusion | 27.0 (24.32) | 25.2 (21.40)
  CFB at 12-hour Follow-up | 0.0 (4.16) | 1.2 (2.94)

26. Primary Outcome: Stage 2: Absolute Values of Serum Chemistry Parameter - Gamma Glutamyl Transferase Levels
Description: Serum chemistry parameters included alanine aminotransferase, aspartate aminotransferase, gamma glutamyl transferase, sodium, potassium, calcium, chloride, bicarbonate, protein, glucose, lactate dehydrogenase, cholesterol, triglycerides, albumin, bilirubin, creatinine, blood urea nitrogen, alkaline phosphatase, creatinine kinase, phosphate, and urate. Absolute values for gamma glutamyl transferase levels are reported in this outcome measure.
Time Frame: Stage 2: Any day in Screening period (Day -7 up to Day -1) and any day in 7-day follow up
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: u/L
Arm/Group | Stage 2: SAGE-547
Number analyzed (Participants) | 17
u/L
  Any Day in Screening Period (Day -7 up to Day -1) | 26.8 (21.72)
  Any Day in 7-day Follow-up | 28.3 (19.65)

27. Primary Outcome: Stage 1: Change From Baseline in Serum Chemistry Parameter - Sodium Levels
Description: Serum chemistry parameters included alanine aminotransferase, aspartate aminotransferase, gamma glutamyl transferase, sodium, potassium, calcium, chloride, bicarbonate, protein, glucose, lactate dehydrogenase, cholesterol, triglycerides, albumin, bilirubin, creatinine, blood urea nitrogen, alkaline phosphatase, creatinine kinase, phosphate, and urate. CFB in sodium levels is reported in this outcome measure. Baseline is defined as the pre-infusion value in each period/stage.
Time Frame: as for outcome 21
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: millimoles per liter (mmol/L)
Arm/Group | Stage 1: SAGE-547 | Stage 1: Placebo
Number analyzed (Participants) | 25 | 25
millimoles per liter (mmol/L)
  Pre-infusion | 140.4 (2.38) | 140.2 (2.35)
  CFB at 12-hour Follow-up | -0.2 (2.19) | -0.6 (3.28)

28. Primary Outcome: Stage 2: Absolute Values of Serum Chemistry Parameter - Sodium Levels
Description: Serum chemistry parameters included alanine aminotransferase, aspartate aminotransferase, gamma glutamyl transferase, sodium, potassium, calcium, chloride, bicarbonate, protein, glucose, lactate dehydrogenase, cholesterol, triglycerides, albumin, bilirubin, creatinine, blood urea nitrogen, alkaline phosphatase, creatinine kinase, phosphate, and urate. Absolute values for sodium levels are reported in this outcome measure.
Time Frame: Stage 2: Any day in Screening period (Day -7 up to Day -1) and any day in 7-day follow up
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Stage 2: SAGE-547
Number analyzed (Participants) | 17
mmol/L
  Any Day in Screening Period (Day -7 up to Day -1) | 139.4 (2.18)
  Any Day in 7-day Follow-up | 139.4 (1.91)

29. Primary Outcome: Stage 1: Change From Baseline in Serum Chemistry Parameter - Potassium Levels
Description: Serum chemistry parameters included alanine aminotransferase, aspartate aminotransferase, gamma glutamyl transferase, sodium, potassium, calcium, chloride, bicarbonate, protein, glucose, lactate dehydrogenase, cholesterol, triglycerides, albumin, bilirubin, creatinine, blood urea nitrogen, alkaline phosphatase, creatinine kinase, phosphate, and urate. CFB in potassium levels is reported in this outcome measure. Baseline is defined as the pre-infusion value in each period/stage.
Time Frame: as for outcome 21
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Stage 1: SAGE-547 | Stage 1: Placebo
Number analyzed (Participants) | 25 | 25
mmol/L
  Pre-infusion | 4.18 (0.273) | 4.17 (0.301)
  CFB at 12-hour Follow-up | -0.00 (0.301) | 0.10 (0.335)

30. Primary Outcome: Stage 2: Absolute Values of Serum Chemistry Parameter - Potassium Levels
Description: Serum chemistry parameters included alanine aminotransferase, aspartate aminotransferase, gamma glutamyl transferase, sodium, potassium, calcium, chloride, bicarbonate, protein, glucose, lactate dehydrogenase, cholesterol, triglycerides, albumin, bilirubin, creatinine, blood urea nitrogen, alkaline phosphatase, creatinine kinase, phosphate, and urate. Absolute values for potassium levels are reported in this outcome measure.
Time Frame: Stage 2: Any day in Screening period (Day -7 up to Day -1) and any day in 7-day follow up
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Stage 2: SAGE-547
Number analyzed (Participants) | 17
mmol/L
  Any Day in Screening Period (Day -7 up to Day -1) | 4.36 (0.232)
  Any Day in 7-day Follow-up | 4.42 (0.268)

31. Primary Outcome: Stage 1: Change From Baseline in Serum Chemistry Parameter - Calcium Levels
Description: Serum chemistry parameters included alanine aminotransferase, aspartate aminotransferase, gamma glutamyl transferase, sodium, potassium, calcium, chloride, bicarbonate, protein, glucose, lactate dehydrogenase, cholesterol, triglycerides, albumin, bilirubin, creatinine, blood urea nitrogen, alkaline phosphatase, creatinine kinase, phosphate, and urate. CFB in calcium levels is reported in this outcome measure. Baseline is defined as the pre-infusion value in each period/stage.
Time Frame: as for outcome 21
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: milligrams per deciliter (mg/dL)
Arm/Group | Stage 1: SAGE-547 | Stage 1: Placebo
Number analyzed (Participants) | 25 | 25
milligrams per deciliter (mg/dL)
  Pre-infusion | 9.07 (0.366) | 9.08 (0.376)
  CFB at 12-hour Follow-up | -0.11 (0.492) | -0.12 (0.393)

32. Primary Outcome: Stage 2: Absolute Values of Serum Chemistry Parameter - Calcium Levels
Description: Serum chemistry parameters included alanine aminotransferase, aspartate aminotransferase, gamma glutamyl transferase, sodium, potassium, calcium, chloride, bicarbonate, protein, glucose, lactate dehydrogenase, cholesterol, triglycerides, albumin, bilirubin, creatinine, blood urea nitrogen, alkaline phosphatase, creatinine kinase, phosphate, and urate. Absolute values for calcium levels are reported in this outcome measure.
Time Frame: Stage 2: Any day in Screening period (Day -7 up to Day -1) and any day in 7-day follow up
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Stage 2: SAGE-547
Number analyzed (Participants) | 17
mg/dL
  Any Day in Screening Period (Day -7 up to Day -1) | 9.19 (0.302)
  Any Day in 7-day Follow-up | 9.12 (0.268)

33. Primary Outcome: Stage 1: Change From Baseline in Serum Chemistry Parameter - Chloride Levels
Description: Serum chemistry parameters included alanine aminotransferase, aspartate aminotransferase, gamma glutamyl transferase, sodium, potassium, calcium, chloride, bicarbonate, protein, glucose, lactate dehydrogenase, cholesterol, triglycerides, albumin, bilirubin, creatinine, blood urea nitrogen, alkaline phosphatase, creatinine kinase, phosphate, and urate. CFB in chloride levels is reported in this outcome measure. Baseline is defined as the pre-infusion value in each period/stage.
Time Frame: as for outcome 21
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Stage 1: SAGE-547 | Stage 1: Placebo
Number analyzed (Participants) | 25 | 25
mmol/L
  Pre-infusion | 106.4 (3.34) | 105.8 (3.00)
  CFB at 12-hour Follow-up | -0.2 (2.54) | -0.2 (2.00)

34. Primary Outcome: Stage 2: Absolute Values of Serum Chemistry Parameter - Chloride Levels
Description: Serum chemistry parameters included alanine aminotransferase, aspartate aminotransferase, gamma glutamyl transferase, sodium, potassium, calcium, chloride, bicarbonate, protein, glucose, lactate dehydrogenase, cholesterol, triglycerides, albumin, bilirubin, creatinine, blood urea nitrogen, alkaline phosphatase, creatinine kinase, phosphate, and urate. Absolute values for chloride levels are reported in this outcome measure.
Time Frame: Stage 2: Any day in Screening period (Day -7 up to Day -1) and any day in 7-day follow up
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Stage 2: SAGE-547
Number analyzed (Participants) | 17
mmol/L
  Any Day in Screening Period (Day -7 up to Day -1) | 103.8 (2.79)
  Any Day in 7-day Follow-up | 104.2 (2.54)

35. Primary Outcome: Stage 1: Change From Baseline in Serum Chemistry Parameter - Bicarbonate Levels
Description: Serum chemistry parameters included alanine aminotransferase, aspartate aminotransferase, gamma glutamyl transferase, sodium, potassium, calcium, chloride, bicarbonate, protein, glucose, lactate dehydrogenase, cholesterol, triglycerides, albumin, bilirubin, creatinine, blood urea nitrogen, alkaline phosphatase, creatinine kinase, phosphate, and urate. CFB in bicarbonate levels is reported in this outcome measure. Baseline is defined as the pre-infusion value in each period/stage.
Time Frame: as for outcome 21
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Stage 1: SAGE-547 | Stage 1: Placebo
Number analyzed (Participants) | 25 | 25
mmol/L
  Pre-infusion | 25.6 (3.47) | 25.6 (2.87)
  CFB at 12-hour Follow-up | -0.4 (2.71) | -0.7 (2.95)

36. Primary Outcome: Stage 2: Absolute Values of Serum Chemistry Parameter - Bicarbonate Levels
Description: Serum chemistry parameters included alanine aminotransferase, aspartate aminotransferase, gamma glutamyl transferase, sodium, potassium, calcium, chloride, bicarbonate, protein, glucose, lactate dehydrogenase, cholesterol, triglycerides, albumin, bilirubin, creatinine, blood urea nitrogen, alkaline phosphatase, creatinine kinase, phosphate, and urate. Absolute values for bicarbonate levels are reported in this outcome measure.
Time Frame: Stage 2: Any day in Screening period (Day -7 up to Day -1) and any day in 7-day follow up
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Stage 2: SAGE-547
Number analyzed (Participants) | 17
mmol/L
  Any Day in Screening Period (Day -7 up to Day -1) | 26.6 (3.91)
  Any Day in 7-day Follow-up | 26.3 (3.60)

37. Primary Outcome: Stage 1: Change From Baseline in Serum Chemistry Parameter - Protein Levels
Description: Serum chemistry parameters included alanine aminotransferase, aspartate aminotransferase, gamma glutamyl transferase, sodium, potassium, calcium, chloride, bicarbonate, protein, glucose, lactate dehydrogenase, cholesterol, triglycerides, albumin, bilirubin, creatinine, blood urea nitrogen, alkaline phosphatase, creatinine kinase, phosphate, and urate. CFB in protein levels is reported in this outcome measure. Baseline is defined as the pre-infusion value in each period/stage.
Time Frame: as for outcome 21
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: grams per deciliter (g/dL)
Arm/Group | Stage 1: SAGE-547 | Stage 1: Placebo
Number analyzed (Participants) | 25 | 25
grams per deciliter (g/dL)
  Pre-infusion | 6.70 (0.452) | 6.66 (0.390)
  CFB at 12-hour Follow-up | -0.08 (0.456) | 0.05 (0.366)

38. Primary Outcome: Stage 2: Absolute Values of Serum Chemistry Parameter - Protein Levels
Description: Serum chemistry parameters included alanine aminotransferase, aspartate aminotransferase, gamma glutamyl transferase, sodium, potassium, calcium, chloride, bicarbonate, protein, glucose, lactate dehydrogenase, cholesterol, triglycerides, albumin, bilirubin, creatinine, blood urea nitrogen, alkaline phosphatase, creatinine kinase, phosphate, and urate. Absolute values for protein levels are reported in this outcome measure.
Time Frame: Stage 2: Any day in Screening period (Day -7 up to Day -1) and any day in 7-day follow up
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Stage 2: SAGE-547
Number analyzed (Participants) | 17
g/dL
  Any Day in Screening Period (Day -7 up to Day -1) | 7.05 (0.403)
  Any Day in 7-day Follow-up | 6.80 (0.417)

39. Primary Outcome: Stage 1: Change From Baseline in Serum Chemistry Parameter - Glucose Levels
Description: Serum chemistry parameters included alanine aminotransferase, aspartate aminotransferase, gamma glutamyl transferase, sodium, potassium, calcium, chloride, bicarbonate, protein, glucose, lactate dehydrogenase, cholesterol, triglycerides, albumin, bilirubin, creatinine, blood urea nitrogen, alkaline phosphatase, creatinine kinase, phosphate, and urate. CFB in glucose levels is reported in this outcome measure. Baseline is defined as the pre-infusion value in each period/stage.
Time Frame: as for outcome 21
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Stage 1: SAGE-547 | Stage 1: Placebo
Number analyzed (Participants) | 25 | 25
mg/dL
  Pre-infusion | 108.0 (34.29) | 95.4 (17.21)
  CFB at 12-hour Follow-up | 0.0 (38.89) | 19.6 (52.94)

40. Primary Outcome: Stage 2: Absolute Values of Serum Chemistry Parameter - Glucose Levels
Description: Serum chemistry parameters included alanine aminotransferase, aspartate aminotransferase, gamma glutamyl transferase, sodium, potassium, calcium, chloride, bicarbonate, protein, glucose, lactate dehydrogenase, cholesterol, triglycerides, albumin, bilirubin, creatinine, blood urea nitrogen, alkaline phosphatase, creatinine kinase, phosphate, and urate. Absolute values for glucose levels are reported in this outcome measure.
Time Frame: Stage 2: Any day in Screening period (Day -7 up to Day -1) and any day in 7-day follow up
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Stage 2: SAGE-547
Number analyzed (Participants) | 17
mg/dL
  Any Day in Screening Period (Day -7 up to Day -1) | 108.1 (60.88)
  Any Day in 7-day Follow-up | 112.8 (71.74)

41. Primary Outcome: Stage 1: Change From Baseline in Serum Chemistry Parameter - Lactate Dehydrogenase Levels
Description: Serum chemistry parameters included alanine aminotransferase, aspartate aminotransferase, gamma glutamyl transferase, sodium, potassium, calcium, chloride, bicarbonate, protein, glucose, lactate dehydrogenase, cholesterol, triglycerides, albumin, bilirubin, creatinine, blood urea nitrogen, alkaline phosphatase, creatinine kinase, phosphate, and urate. CFB in lactate dehydrogenase levels is reported in this outcome measure. Baseline is defined as the pre-infusion value in each period/stage.
Time Frame: as for outcome 21
Population: Safety population included all participants admitted into the inpatient unit who met all eligibility criteria, signed an informed consent, and who began infusion with SAGE-547 or placebo in Treatment Period 1 of Stage 1. Overall number of participants analyzed = Number of participants analyzed in this outcome measure. Number analyzed = Number of participants with data available at the specific time point.
Measure: Mean (Standard Deviation); unit: u/L
Arm/Group | Stage 1: SAGE-547 | Stage 1: Placebo
Number analyzed (Participants) | 15 | 14
u/L
  Pre-infusion | 167.9 (32.75) | 153.1 (29.87)
  CFB at 12-hour Follow-up: number analyzed (Participants) | 13 | 13
  CFB at 12-hour Follow-up | -16.6 (15.59) | -0.8 (17.57)

42. Primary Outcome: Stage 2: Absolute Values of Serum Chemistry Parameter - Lactate Dehydrogenase Levels
Description: Serum chemistry parameters included alanine aminotransferase, aspartate aminotransferase, gamma glutamyl transferase, sodium, potassium, calcium, chloride, bicarbonate, protein, glucose, lactate dehydrogenase, cholesterol, triglycerides, albumin, bilirubin, creatinine, blood urea nitrogen, alkaline phosphatase, creatinine kinase, phosphate, and urate. Absolute values for lactate dehydrogenase levels are reported in this outcome measure.
Time Frame: Stage 2: Any day in Screening period (Day -7 up to Day -1) and any day in 7-day follow up
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: u/L
Arm/Group | Stage 2: SAGE-547
Number analyzed (Participants) | 17
u/L
  Any Day in Screening Period (Day -7 up to Day -1) | 162.9 (39.06)
  Any Day in 7-day Follow-up | 168.8 (40.97)

43. Primary Outcome: Stage 1: Change From Baseline in Serum Chemistry Parameter - Cholesterol Levels
Description: Serum chemistry parameters included alanine aminotransferase, aspartate aminotransferase, gamma glutamyl transferase, sodium, potassium, calcium, chloride, bicarbonate, protein, glucose, lactate dehydrogenase, cholesterol, triglycerides, albumin, bilirubin, creatinine, blood urea nitrogen, alkaline phosphatase, creatinine kinase, phosphate, and urate. CFB in cholesterol levels is reported in this outcome measure. Baseline is defined as the pre-infusion value in each period/stage.
Time Frame: as for outcome 21
Population: as for outcome 41
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Stage 1: SAGE-547 | Stage 1: Placebo
Number analyzed (Participants) | 23 | 23
mg/dL
  Pre-infusion | 183.0 (32.77) | 183.4 (24.63)
  CFB at 12-hour Follow-up: number analyzed (Participants) | 21 | 21
  CFB at 12-hour Follow-up | 0.4 (14.01) | 2.1 (20.84)

44. Primary Outcome: Stage 2: Absolute Values of Serum Chemistry Parameter - Cholesterol Level
Description: Serum chemistry parameters included alanine aminotransferase, aspartate aminotransferase, gamma glutamyl transferase, sodium, potassium, calcium, chloride, bicarbonate, protein, glucose, lactate dehydrogenase, cholesterol, triglycerides, albumin, bilirubin, creatinine, blood urea nitrogen, alkaline phosphatase, creatinine kinase, phosphate, and urate. Absolute values for cholesterol levels are reported in this outcome measure.
Time Frame: Stage 2: Any day in Screening period (Day -7 up to Day -1) and any day in 7-day follow up
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Stage 2: SAGE-547
Number analyzed (Participants) | 17
mg/dL
  Any Day in Screening Period (Day -7 up to Day -1) | 194.6 (39.64)
  Any Day in 7-day Follow-up | 179.7 (33.94)

45. Primary Outcome: Stage 1: Change From Baseline in Serum Chemistry Parameter - Triglyceride Levels
Description: Serum chemistry parameters included alanine aminotransferase, aspartate aminotransferase, gamma glutamyl transferase, sodium, potassium, calcium, chloride, bicarbonate, protein, glucose, lactate dehydrogenase, cholesterol, triglycerides, albumin, bilirubin, creatinine, blood urea nitrogen, alkaline phosphatase, creatinine kinase, phosphate, and urate. CFB in triglyceride levels is reported in this outcome measure. Baseline is defined as the pre-infusion value in each period/stage.
Time Frame: as for outcome 21
Population: as for outcome 41
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Stage 1: SAGE-547 | Stage 1: Placebo
Number analyzed (Participants) | 23 | 23
mg/dL
  Pre-infusion | 166.1 (93.42) | 168.4 (77.72)
  CFB at 12-hour Follow-up: number analyzed (Participants) | 21 | 21
  CFB at 12-hour Follow-up | -19.1 (67.47) | -25.1 (45.41)

46. Primary Outcome: Stage 2: Absolute Values of Serum Chemistry Parameter - Triglyceride Levels
Description: Serum chemistry parameters included alanine aminotransferase, aspartate aminotransferase, gamma glutamyl transferase, sodium, potassium, calcium, chloride, bicarbonate, protein, glucose, lactate dehydrogenase, cholesterol, triglycerides, albumin, bilirubin, creatinine, blood urea nitrogen, alkaline phosphatase, creatinine kinase, phosphate, and urate. Absolute values for triglyceride levels are reported in this outcome measure.
Time Frame: Stage 2: Any day in Screening period (Day -7 up to Day -1) and any day in 7-day follow up
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Stage 2: SAGE-547
Number analyzed (Participants) | 17
mg/dL
  Any Day in Screening Period (Day -7 up to Day -1) | 162.4 (63.59)
  Any Day in 7-day Follow-up | 163.4 (69.94)

47. Primary Outcome: Stage 1: Change From Baseline in Serum Chemistry Parameter - Albumin Levels
Description: Serum chemistry parameters included alanine aminotransferase, aspartate aminotransferase, gamma glutamyl transferase, sodium, potassium, calcium, chloride, bicarbonate, protein, glucose, lactate dehydrogenase, cholesterol, triglycerides, albumin, bilirubin, creatinine, blood urea nitrogen, alkaline phosphatase, creatinine kinase, phosphate, and urate. CFB in albumin levels is reported in this outcome measure. Baseline is defined as the pre-infusion value in each period/stage.
Time Frame: as for outcome 21
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Stage 1: SAGE-547 | Stage 1: Placebo
Number analyzed (Participants) | 25 | 25
g/dL
  Pre-infusion | 3.94 (0.260) | 3.95 (0.315)
  CFB at 12-hour Follow-up | -0.06 (0.314) | -0.01 (0.276)

48. Primary Outcome: Stage 2: Absolute Values of Serum Chemistry Parameter - Albumin Levels
Description: Serum chemistry parameters included alanine aminotransferase, aspartate aminotransferase, gamma glutamyl transferase, sodium, potassium, calcium, chloride, bicarbonate, protein, glucose, lactate dehydrogenase, cholesterol, triglycerides, albumin, bilirubin, creatinine, blood urea nitrogen, alkaline phosphatase, creatinine kinase, phosphate, and urate. Absolute values for albumin levels are reported in this outcome measure.
Time Frame: Stage 2: Any day in Screening period (Day -7 up to Day -1) and any day in 7-day follow up
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Stage 2: SAGE-547
Number analyzed (Participants) | 17
g/dL
  Any Day in Screening Period (Day -7 up to Day -1) | 4.03 (0.331)
  Any Day in 7-day Follow-up | 3.92 (0.299)

49. Primary Outcome: Stage 1: Change From Baseline in Serum Chemistry Parameter - Bilirubin Levels
Description: Serum chemistry parameters included alanine aminotransferase, aspartate aminotransferase, gamma glutamyl transferase, sodium, potassium, calcium, chloride, bicarbonate, protein, glucose, lactate dehydrogenase, cholesterol, triglycerides, albumin, bilirubin, creatinine, blood urea nitrogen, alkaline phosphatase, creatinine kinase, phosphate, and urate. CFB in bilirubin levels is reported in this outcome measure. Baseline is defined as the pre-infusion value in each period/stage.
Time Frame: as for outcome 21
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Stage 1: SAGE-547 | Stage 1: Placebo
Number analyzed (Participants) | 25 | 25
mg/dL
  Pre-infusion | 0.44 (0.231) | 0.47 (0.313)
  CFB at 12-hour Follow-up | 0.04 (0.144) | 0.09 (0.127)

50. Primary Outcome: Stage 2: Absolute Values of Serum Chemistry Parameter - Bilirubin Levels
Description: Serum chemistry parameters included alanine aminotransferase, aspartate aminotransferase, gamma glutamyl transferase, sodium, potassium, calcium, chloride, bicarbonate, protein, glucose, lactate dehydrogenase, cholesterol, triglycerides, albumin, bilirubin, creatinine, blood urea nitrogen, alkaline phosphatase, creatinine kinase, phosphate, and urate. Absolute values for bilirubin levels are reported in this outcome measure.
Time Frame: Stage 2: Any day in Screening period (Day -7 up to Day -1) and any day in 7-day follow up
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Stage 2: SAGE-547
Number analyzed (Participants) | 17
mg/dL
  Any Day in Screening Period (Day -7 up to Day -1) | 0.58 (0.354)
  Any Day in 7-day Follow-up | 0.57 (0.463)

51. Primary Outcome: Stage 1: Change From Baseline in Serum Chemistry Parameter - Creatinine Levels
Description: Serum chemistry parameters included alanine aminotransferase, aspartate aminotransferase, gamma glutamyl transferase, sodium, potassium, calcium, chloride, bicarbonate, protein, glucose, lactate dehydrogenase, cholesterol, triglycerides, albumin, bilirubin, creatinine, blood urea nitrogen, alkaline phosphatase, creatinine kinase, phosphate, and urate. CFB in creatinine levels is reported in this outcome measure. Baseline is defined as the pre-infusion value in each period/stage.
Time Frame: as for outcome 21
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Stage 1: SAGE-547 | Stage 1: Placebo
Number analyzed (Participants) | 25 | 25
mg/dL
  Pre-infusion | 0.940 (0.2480) | 0.951 (0.2912)
  CFB at 12-hour Follow-up | -0.07 (0.104) | -0.09 (0.128)

52. Primary Outcome: Stage 2: Absolute Values of Serum Chemistry Parameter - Creatinine Levels
Description: Serum chemistry parameters included alanine aminotransferase, aspartate aminotransferase, gamma glutamyl transferase, sodium, potassium, calcium, chloride, bicarbonate, protein, glucose, lactate dehydrogenase, cholesterol, triglycerides, albumin, bilirubin, creatinine, blood urea nitrogen, alkaline phosphatase, creatinine kinase, phosphate, and urate. Absolute values for creatinine levels are reported in this outcome measure.
Time Frame: Stage 2: Any day in Screening period (Day -7 up to Day -1) and any day in 7-day follow up
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Stage 2: SAGE-547
Number analyzed (Participants) | 17
mg/dL
  Any Day in Screening Period (Day -7 up to Day -1) | 0.872 (0.2302)
  Any Day in 7-day Follow-up | 0.912 (0.2234)

53. Primary Outcome: Stage 1: Change From Baseline in Serum Chemistry Parameter - Blood Urea Nitrogen Levels
Description: Serum chemistry parameters included alanine aminotransferase, aspartate aminotransferase, gamma glutamyl transferase, sodium, potassium, calcium, chloride, bicarbonate, protein, glucose, lactate dehydrogenase, cholesterol, triglycerides, albumin, bilirubin, creatinine, blood urea nitrogen, alkaline phosphatase, creatinine kinase, phosphate, and urate. CFB in blood urea nitrogen levels is reported in this outcome measure. Baseline is defined as the pre-infusion value in each period/stage.
Time Frame: as for outcome 21
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Stage 1: SAGE-547 | Stage 1: Placebo
Number analyzed (Participants) | 25 | 25
mg/dL
  Pre-infusion | 18.1 (4.60) | 17.9 (5.73)
  CFB at 12-hour Follow-up | -0.4 (4.36) | -0.3 (3.08)

54. Primary Outcome: Stage 2: Absolute Values of Serum Chemistry Parameter - Blood Urea Nitrogen Levels
Description: Serum chemistry parameters included alanine aminotransferase, aspartate aminotransferase, gamma glutamyl transferase, sodium, potassium, calcium, chloride, bicarbonate, protein, glucose, lactate dehydrogenase, cholesterol, triglycerides, albumin, bilirubin, creatinine, blood urea nitrogen, alkaline phosphatase, creatinine kinase, phosphate, and urate. Absolute values for blood urea nitrogen levels are reported in this outcome measure.
Time Frame: Stage 2: Any day in Screening period (Day -7 up to Day -1) and any day in 7-day follow up
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Stage 2: SAGE-547
Number analyzed (Participants) | 17
mg/dL
  Any Day in Screening Period (Day -7 up to Day -1) | 17.3 (4.31)
  Any Day in 7-day Follow-up | 16.6 (3.37)

55. Primary Outcome: Stage 1: Change From Baseline in Serum Chemistry Parameter - Alkaline Phosphatase Levels
Description: Serum chemistry parameters included alanine aminotransferase, aspartate aminotransferase, gamma glutamyl transferase, sodium, potassium, calcium, chloride, bicarbonate, protein, glucose, lactate dehydrogenase, cholesterol, triglycerides, albumin, bilirubin, creatinine, blood urea nitrogen, alkaline phosphatase, creatinine kinase, phosphate, and urate. CFB in alkaline phosphatase levels is reported in this outcome measure. Baseline is defined as the pre-infusion value in each period/stage.
Time Frame: as for outcome 21
Population: Safety population included all participants admitted into the inpatient unit who met all eligibility criteria, signed an informed consent, and who began infusion with SAGE-547 or placebo in Treatment Period 1 of Stage 1. Overall number of participants analyzed = Number of participants analyzed in this outcome measure.
Measure: Mean (Standard Deviation); unit: u/L
Arm/Group | Stage 1: SAGE-547 | Stage 1: Placebo
Number analyzed (Participants) | 23 | 23
u/L
  Pre-infusion | 69.1 (13.97) | 67.1 (13.58)
  CFB at 12-hour Follow-up | -2.4 (5.37) | -0.4 (6.83)

56. Primary Outcome: Stage 2: Absolute Values of Serum Chemistry Parameter - Alkaline Phosphatase Levels
Description: Serum chemistry parameters included alanine aminotransferase, aspartate aminotransferase, gamma glutamyl transferase, sodium, potassium, calcium, chloride, bicarbonate, protein, glucose, lactate dehydrogenase, cholesterol, triglycerides, albumin, bilirubin, creatinine, blood urea nitrogen, alkaline phosphatase, creatinine kinase, phosphate, and urate. Absolute values for alkaline phosphatase levels are reported in this outcome measure.
Time Frame: Stage 2: Any day in Screening period (Day -7 up to Day -1) and any day in 7-day follow up
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: u/L
Arm/Group | Stage 2: SAGE-547
Number analyzed (Participants) | 17
u/L
  Any Day in Screening Period (Day -7 up to Day -1) | 71.1 (13.99)
  Any Day in 7-day Follow-up | 71.4 (14.33)

57. Primary Outcome: Stage 1: Change From Baseline in Serum Chemistry Parameter - Creatine Kinase Levels
Description: Serum chemistry parameters included alanine aminotransferase, aspartate aminotransferase, gamma glutamyl transferase, sodium, potassium, calcium, chloride, bicarbonate, protein, glucose, lactate dehydrogenase, cholesterol, triglycerides, albumin, bilirubin, creatinine, blood urea nitrogen, alkaline phosphatase, creatinine kinase, phosphate, and urate. CFB in creatinine kinase levels is reported in this outcome measure. Baseline is defined as the pre-infusion value in each period/stage.
Time Frame: as for outcome 21
Population: as for outcome 55
Measure: Mean (Standard Deviation); unit: u/L
Arm/Group | Stage 1: SAGE-547 | Stage 1: Placebo
Number analyzed (Participants) | 23 | 21
u/L
  Pre-infusion | 100.5 (71.25) | 124.0 (188.98)
  CFB at 12-hour Follow-up | -20.6 (25.57) | -36.2 (90.71)

58. Primary Outcome: Stage 2: Absolute Values of Serum Chemistry Parameter - Creatine Kinase Levels
Description: Serum chemistry parameters included alanine aminotransferase, aspartate aminotransferase, gamma glutamyl transferase, sodium, potassium, calcium, chloride, bicarbonate, protein, glucose, lactate dehydrogenase, cholesterol, triglycerides, albumin, bilirubin, creatinine, blood urea nitrogen, alkaline phosphatase, creatinine kinase, phosphate, and urate. Absolute values for creatinine kinase levels are reported in this outcome measure.
Time Frame: Stage 2: Any day in Screening period (Day -7 up to Day -1) and any day in 7-day follow up
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: u/L
Arm/Group | Stage 2: SAGE-547
Number analyzed (Participants) | 17
u/L
  Any Day in Screening Period (Day -7 up to Day -1) | 83.9 (32.51)
  Any Day in 7-day Follow-up | 85.9 (44.45)

59. Primary Outcome: Stage 1: Change From Baseline in Serum Chemistry Parameter - Phosphate Levels
Description: Serum chemistry parameters included alanine aminotransferase, aspartate aminotransferase, gamma glutamyl transferase, sodium, potassium, calcium, chloride, bicarbonate, protein, glucose, lactate dehydrogenase, cholesterol, triglycerides, albumin, bilirubin, creatinine, blood urea nitrogen, alkaline phosphatase, creatinine kinase, phosphate, and urate. CFB in phosphate levels is reported in this outcome measure. Baseline is defined as the pre-infusion value in each period/stage.
Time Frame: as for outcome 21
Population: Safety population included all participants admitted into the inpatient unit who met all eligibility criteria, signed an informed consent, and who began infusion with SAGE-547 or placebo in Treatment Period 1 of Stage 1. Number analyzed = Number of participants with data available at the specific time point.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Stage 1: SAGE-547 | Stage 1: Placebo
Number analyzed (Participants) | 25 | 25
mg/dL
  Pre-infusion: number analyzed (Participants) | 22 | 23
  Pre-infusion | 3.58 (0.468) | 3.52 (0.551)
  CFB at 12-hour Follow-up: number analyzed (Participants) | 23 | 23
  CFB at 12-hour Follow-up | -0.16 (0.481) | -0.17 (0.581)

60. Primary Outcome: Stage 2: Absolute Values of Serum Chemistry Parameter - Phosphate Levels
Description: Serum chemistry parameters included alanine aminotransferase, aspartate aminotransferase, gamma glutamyl transferase, sodium, potassium, calcium, chloride, bicarbonate, protein, glucose, lactate dehydrogenase, cholesterol, triglycerides, albumin, bilirubin, creatinine, blood urea nitrogen, alkaline phosphatase, creatinine kinase, phosphate, and urate. Absolute values for phosphate levels are reported in this outcome measure.
Time Frame: Stage 2: Any day in Screening period (Day -7 up to Day -1) and any day in 7-day follow up
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Stage 2: SAGE-547
Number analyzed (Participants) | 17
mg/dL
  Any Day in Screening Period (Day -7 up to Day -1) | 3.36 (0.436)
  Any Day in 7-day Follow-up | 3.23 (0.461)

61. Primary Outcome: Stage 1: Change From Baseline in Serum Chemistry Parameter - Urate Levels
Description: Serum chemistry parameters included alanine aminotransferase, aspartate aminotransferase, gamma glutamyl transferase, sodium, potassium, calcium, chloride, bicarbonate, protein, glucose, lactate dehydrogenase, cholesterol, triglycerides, albumin, bilirubin, creatinine, blood urea nitrogen, alkaline phosphatase, creatinine kinase, phosphate, and urate. CFB in urate levels is reported in this outcome measure. Baseline is defined as the pre-infusion value in each period/stage.
Time Frame: as for outcome 21
Population: as for outcome 55
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Stage 1: SAGE-547 | Stage 1: Placebo
Number analyzed (Participants) | 23 | 23
mg/dL
  Pre-infusion | 4.53 (1.249) | 4.71 (1.366)
  CFB at 12-hour Follow-up | 0.05 (0.532) | -0.04 (0.317)

62. Primary Outcome: Stage 2: Absolute Values of Serum Chemistry Parameter - Urate Levels
Description: Serum chemistry parameters included alanine aminotransferase, aspartate aminotransferase, gamma glutamyl transferase, sodium, potassium, calcium, chloride, bicarbonate, protein, glucose, lactate dehydrogenase, cholesterol, triglycerides, albumin, bilirubin, creatinine, blood urea nitrogen, alkaline phosphatase, creatinine kinase, phosphate, and urate. Absolute values for urate levels are reported in this outcome measure.
Time Frame: Stage 2: Any day in Screening period (Day -7 up to Day -1) and any day in 7-day follow up
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Stage 2: SAGE-547
Number analyzed (Participants) | 17
mg/dL
  Any Day in Screening Period (Day -7 up to Day -1) | 4.66 (1.169)
  Any Day in 7-day Follow-up | 4.84 (1.183)

63. Primary Outcome: Stage 1: Change From Baseline in Hematology Parameter - Hemoglobin Levels
Description: Hematology parameters included hemoglobin, hematocrit, platelets, erythrocytes, neutrophils, basophils, eosinophils, monocytes, lymphocytes, leukocytes, erythrocytes mean corpuscular volume, and mean cell hemoglobin. CFB in hemoglobin levels is reported in this outcome measure. Baseline is defined as the pre-infusion value in each period/stage.
Time Frame: as for outcome 21
Population: as for outcome 59
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Stage 1: SAGE-547 | Stage 1: Placebo
Number analyzed (Participants) | 25 | 25
g/dL
  Pre-infusion | 13.56 (1.276) | 13.63 (1.179)
  CFB at 12-hours Follow-up: number analyzed (Participants) | 25 | 24
  CFB at 12-hours Follow-up | 0.34 (0.733) | 0.28 (0.768)

64. Primary Outcome: Stage 2: Absolute Values of Hematology Parameter - Hemoglobin Levels
Description: Hematology parameters included hemoglobin, hematocrit, platelets, erythrocytes, neutrophils, basophils, eosinophils, monocytes, lymphocytes, leukocytes, erythrocytes mean corpuscular volume, and mean cell hemoglobin. Absolute values for hemoglobin levels are reported in this outcome measure.
Time Frame: Stage 2: Any day in Screening period (Day -7 up to Day -1) and any day in 7-day follow up
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Stage 2: SAGE-547
Number analyzed (Participants) | 17
g/dL
  Any Day in Screening Period (Day -7 up to Day -1) | 14.74 (1.419)
  Any Day in 7-day Follow-up | 14.11 (1.684)

65. Primary Outcome: Stage 1: Change From Baseline in Hematology Parameter - Hematocrit Levels
Description: Hematology parameters included hemoglobin, hematocrit, platelets, erythrocytes, neutrophils, basophils, eosinophils, monocytes, lymphocytes, leukocytes, erythrocytes mean corpuscular volume, and mean cell hemoglobin. CFB in hematocrit levels is reported in this outcome measure. Baseline is defined as the pre-infusion value in each period/stage.
Time Frame: as for outcome 21
Population: as for outcome 59
Measure: Mean (Standard Deviation); unit: percentage of cells
Arm/Group | Stage 1: SAGE-547 | Stage 1: Placebo
Number analyzed (Participants) | 25 | 25
percentage of cells
  Pre-infusion | 40.66 (3.463) | 40.97 (3.453)
  CFB at 12-hours Follow-up: number analyzed (Participants) | 25 | 24
  CFB at 12-hours Follow-up | 1.02 (2.013) | 0.67 (2.494)

66. Primary Outcome: Stage 2: Absolute Values of Hematology Parameter - Hematocrit Levels
Description: Hematology parameters included hemoglobin, hematocrit, platelets, erythrocytes, neutrophils, basophils, eosinophils, monocytes, lymphocytes, leukocytes, erythrocytes mean corpuscular volume, and mean cell hemoglobin. Absolute values for hematocrit levels are reported in this outcome measure.
Time Frame: Stage 2: Any day in Screening period (Day -7 up to Day -1) and any day in 7-day follow up
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage of cells
Arm/Group | Stage 2: SAGE-547
Number analyzed (Participants) | 17
percentage of cells
  Any Day in Screening Period (Day -7 up to Day -1) | 45.04 (4.230)
  Any Day in 7-day Follow-up | 43.28 (5.128)

67. Primary Outcome: Stage 1: Change From Baseline in Hematology Parameter - Platelet Levels
Description: Hematology parameters included hemoglobin, hematocrit, platelets, erythrocytes, neutrophils, basophils, eosinophils, monocytes, lymphocytes, leukocytes, erythrocytes mean corpuscular volume, and mean cell hemoglobin. CFB in platelet levels is reported in this outcome measure. Baseline is defined as the pre-infusion value in each period/stage.
Time Frame: as for outcome 21
Population: as for outcome 59
Measure: Mean (Standard Deviation); unit: 10^3 cells per microliter(10^3 cells/μL)
Arm/Group | Stage 1: SAGE-547 | Stage 1: Placebo
Number analyzed (Participants) | 25 | 25
10^3 cells per microliter(10^3 cells/μL)
  Pre-infusion | 212.5 (40.56) | 218.8 (48.31)
  CFB at 12-hours Follow-up: number analyzed (Participants) | 25 | 24
  CFB at 12-hours Follow-up | -11.7 (45.02) | -7.1 (37.11)

68. Primary Outcome: Stage 2: Absolute Values of Hematology Parameter - Platelet Levels
Description: Hematology parameters included hemoglobin, hematocrit, platelets, erythrocytes, neutrophils, basophils, eosinophils, monocytes, lymphocytes, leukocytes, erythrocytes mean corpuscular volume, and mean cell hemoglobin. Absolute values for platelet levels are reported in this outcome measure.
Time Frame: Stage 2: Any day in Screening period (Day -7 up to Day -1) and any day in 7-day follow up
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: 10^3 cells/μL
Arm/Group | Stage 2: SAGE-547
Number analyzed (Participants) | 17
10^3 cells/μL
  Any Day in Screening Period (Day -7 up to Day -1) | 233.8 (48.03)
  Any Day in 7-day Follow-up | 230.5 (45.93)

69. Primary Outcome: Stage 1: Change From Baseline in Hematology Parameter - Erythrocyte Levels
Description: Hematology parameters included hemoglobin, hematocrit, platelets, erythrocytes, neutrophils, basophils, eosinophils, monocytes, lymphocytes, leukocytes, erythrocytes mean corpuscular volume, and mean cell hemoglobin. CFB in erythrocyte levels is reported in this outcome measure. Baseline is defined as the pre-infusion value in each period/stage.
Time Frame: as for outcome 21
Population: as for outcome 59
Measure: Mean (Standard Deviation); unit: 10^6 cells per microliter(10^6 cells/μL)
Arm/Group | Stage 1: SAGE-547 | Stage 1: Placebo
Number analyzed (Participants) | 25 | 25
10^6 cells per microliter(10^6 cells/μL)
  Pre-infusion | 4.437 (0.4032) | 4.474 (0.4119)
  CFB at 12-hours Follow-up: number analyzed (Participants) | 25 | 24
  CFB at 12-hours Follow-up | 0.09 (0.223) | 0.07 (0.271)

70. Primary Outcome: Stage 2: Absolute Values of Hematology Parameter - Erythrocyte Levels
Description: Hematology parameters included hemoglobin, hematocrit, platelets, erythrocytes, neutrophils, basophils, eosinophils, monocytes, lymphocytes, leukocytes, erythrocytes mean corpuscular volume, and mean cell hemoglobin. Absolute values for erythrocyte levels are reported in this outcome measure.
Time Frame: Stage 2: Any day in Screening period (Day -7 up to Day -1) and any day in 7-day follow up
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: 10^6 cells/μL
Arm/Group | Stage 2: SAGE-547
Number analyzed (Participants) | 17
10^6 cells/μL
  Any Day in Screening Period (Day -7 up to Day -1) | 4.925 (0.4173)
  Any Day in 7-day Follow-up | 4.735 (0.5289)

71. Primary Outcome: Stage 1: Change From Baseline in Hematology Parameter - Neutrophil Levels
Description: Hematology parameters included hemoglobin, hematocrit, platelets, erythrocytes, neutrophils, basophils, eosinophils, monocytes, lymphocytes, leukocytes, erythrocytes mean corpuscular volume, and mean cell hemoglobin. CFB in neutrophil levels is reported in this outcome measure. Baseline is defined as the pre-infusion value in each period/stage.
Time Frame: as for outcome 21
Population: as for outcome 55
Measure: Mean (Standard Deviation); unit: 10^3 cells/μL
Arm/Group | Stage 1: SAGE-547 | Stage 1: Placebo
Number analyzed (Participants) | 12 | 12
10^3 cells/μL
  Pre-infusion | 4.510 (1.2311) | 4.781 (1.6007)
  CFB at 12-hours Follow-up | -0.49 (0.941) | -0.66 (1.053)

72. Primary Outcome: Stage 2: Absolute Values of Hematology Parameter - Neutrophil Levels
Description: Hematology parameters included hemoglobin, hematocrit, platelets, erythrocytes, neutrophils, basophils, eosinophils, monocytes, lymphocytes, leukocytes, erythrocytes mean corpuscular volume, and mean cell hemoglobin. Absolute values for neutrophil levels are reported in this outcome measure.
Time Frame: Stage 2: Any day in Screening period (Day -7 up to Day -1) and any day in 7-day follow up
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: 10^3 cells/μL
Arm/Group | Stage 2: SAGE-547
Number analyzed (Participants) | 11
10^3 cells/μL
  Any Day in Screening Period (Day -7 up to Day -1) | 4.049 (0.8958)
  Any Day in 7-day Follow-up: number analyzed (Participants) | 10
  Any Day in 7-day Follow-up | 4.176 (0.8065)

73. Primary Outcome: Stage 1: Change From Baseline in Hematology Parameter - Basophil Levels
Description: Hematology parameters included hemoglobin, hematocrit, platelets, erythrocytes, neutrophils, basophils, eosinophils, monocytes, lymphocytes, leukocytes, erythrocytes mean corpuscular volume, and mean cell hemoglobin. CFB in basophil levels is reported in this outcome measure. Baseline is defined as the pre-infusion value in each period/stage.
Time Frame: as for outcome 21
Population: as for outcome 41
Measure: Mean (Standard Deviation); unit: cells per microliter (cells/μL)
Arm/Group | Stage 1: SAGE-547 | Stage 1: Placebo
Number analyzed (Participants) | 13 | 13
cells per microliter (cells/μL)
  Pre-infusion | 25.4 (15.61) | 27.2 (20.45)
  CFB at 12-hours Follow-up: number analyzed (Participants) | 13 | 12
  CFB at 12-hours Follow-up | 6.4 (17.06) | -8.3 (21.83)

74. Primary Outcome: Stage 2: Absolute Values of Hematology Parameter - Basophil Levels
Description: Hematology parameters included hemoglobin, hematocrit, platelets, erythrocytes, neutrophils, basophils, eosinophils, monocytes, lymphocytes, leukocytes, erythrocytes mean corpuscular volume, and mean cell hemoglobin. Absolute values for basophil levels are reported in this outcome measure.
Time Frame: Stage 2: Any day in Screening period (Day -7 up to Day -1) and any day in 7-day follow up
Population: Participants from safety population, which included all participants admitted into the inpatient unit who met all eligibility criteria, signed an informed consent, and who began infusion with SAGE-547 or placebo in Treatment Period 1, who received study drug in Stage 2. Overall number of participants analyzed = Number of participants analyzed in this outcome measure.
Measure: Mean (Standard Deviation); unit: cells/μL
Arm/Group | Stage 2: SAGE-547
Number analyzed (Participants) | 6
cells/μL
  Any Day in Screening Period (Day -7 up to Day -1) | 35.3 (20.70)
  Any Day in 7-day Follow-up | 45.3 (47.64)

75. Primary Outcome: Stage 1: Change From Baseline in Hematology Parameter - Eosinophil Levels
Description: Hematology parameters included hemoglobin, hematocrit, platelets, erythrocytes, neutrophils, basophils, eosinophils, monocytes, lymphocytes, leukocytes, erythrocytes mean corpuscular volume, and mean cell hemoglobin. CFB in eosinophil levels is reported in this outcome measure. Baseline is defined as the pre-infusion value in each period/stage.
Time Frame: as for outcome 21
Population: as for outcome 41
Measure: Mean (Standard Deviation); unit: cells/μL
Arm/Group | Stage 1: SAGE-547 | Stage 1: Placebo
Number analyzed (Participants) | 13 | 13
cells/μL
  Pre-infusion | 158.8 (77.53) | 140.3 (109.72)
  CFB at 12-hours Follow-up: number analyzed (Participants) | 13 | 12
  CFB at 12-hours Follow-up | 11.5 (45.21) | 42.5 (47.48)

76. Primary Outcome: Stage 2: Absolute Values of Hematology Parameter - Eosinophil Levels
Description: Hematology parameters included hemoglobin, hematocrit, platelets, erythrocytes, neutrophils, basophils, eosinophils, monocytes, lymphocytes, leukocytes, erythrocytes mean corpuscular volume, and mean cell hemoglobin. Absolute values for eosinophil levels are reported in this outcome measure.
Time Frame: Stage 2: Any day in Screening period (Day -7 up to Day -1) and any day in 7-day follow up
Population: as for outcome 74
Measure: Mean (Standard Deviation); unit: cells/μL
Arm/Group | Stage 2: SAGE-547
Number analyzed (Participants) | 6
cells/μL
  Any Day in Screening Period (Day -7 up to Day -1) | 87.2 (40.49)
  Any Day in 7-day Follow-up | 99.8 (75.37)

77. Primary Outcome: Stage 1: Change From Baseline in Hematology Parameter - Monocyte Levels
Description: Hematology parameters included hemoglobin, hematocrit, platelets, erythrocytes, neutrophils, basophils, eosinophils, monocytes, lymphocytes, leukocytes, erythrocytes mean corpuscular volume, and mean cell hemoglobin. CFB in monocyte levels is reported in this outcome measure. Baseline is defined as the pre-infusion value in each period/stage.
Time Frame: as for outcome 21
Population: as for outcome 41
Measure: Mean (Standard Deviation); unit: cells/μL
Arm/Group | Stage 1: SAGE-547 | Stage 1: Placebo
Number analyzed (Participants) | 13 | 13
cells/μL
  Pre-infusion | 480.5 (264.68) | 462.8 (240.92)
  CFB at 12-hours Follow-up: number analyzed (Participants) | 13 | 12
  CFB at 12-hours Follow-up | -22.9 (176.01) | -40.3 (113.21)

78. Primary Outcome: Stage 2: Absolute Values of Hematology Parameter - Monocyte Levels
Description: Hematology parameters included hemoglobin, hematocrit, platelets, erythrocytes, neutrophils, basophils, eosinophils, monocytes, lymphocytes, leukocytes, erythrocytes mean corpuscular volume, and mean cell hemoglobin. Absolute values for monocyte levels are reported in this outcome measure.
Time Frame: Stage 2: Any day in Screening period (Day -7 up to Day -1) and any day in 7-day follow up
Population: as for outcome 74
Measure: Mean (Standard Deviation); unit: cells/μL
Arm/Group | Stage 2: SAGE-547
Number analyzed (Participants) | 6
cells/μL
  Any Day in Screening Period (Day -7 up to Day -1) | 499.8 (190.38)
  Any Day in 7-day Follow-up | 426.7 (133.11)

79. Primary Outcome: Stage 1: Change From Baseline in Hematology Parameter - Lymphocyte Levels
Description: Hematology parameters included hemoglobin, hematocrit, platelets, erythrocytes, neutrophils, basophils, eosinophils, monocytes, lymphocytes, leukocytes, erythrocytes mean corpuscular volume, and mean cell hemoglobin. CFB in lymphocyte levels is reported in this outcome measure. Baseline is defined as the pre-infusion value in each period/stage.
Time Frame: as for outcome 21
Population: as for outcome 41
Measure: Mean (Standard Deviation); unit: cells/μL
Arm/Group | Stage 1: SAGE-547 | Stage 1: Placebo
Number analyzed (Participants) | 13 | 13
cells/μL
  Pre-infusion | 1641.7 (423.63) | 1590.1 (427.61)
  CFB at 12-hours Follow-up: number analyzed (Participants) | 13 | 12
  CFB at 12-hours Follow-up | 176.5 (244.63) | 100.3 (310.99)

80. Primary Outcome: Stage 2: Absolute Values of Hematology Parameter - Lymphocyte Levels
Description: Hematology parameters included hemoglobin, hematocrit, platelets, erythrocytes, neutrophils, basophils, eosinophils, monocytes, lymphocytes, leukocytes, erythrocytes mean corpuscular volume, and mean cell hemoglobin. Absolute values for lymphocyte levels are reported in this outcome measure.
Time Frame: Stage 2: Any day in Screening period (Day -7 up to Day -1) and any day in 7-day follow up
Population: as for outcome 74
Measure: Mean (Standard Deviation); unit: cells/μL
Arm/Group | Stage 2: SAGE-547
Number analyzed (Participants) | 6
cells/μL
  Any Day in Screening Period (Day -7 up to Day -1) | 2080.0 (908.52)
  Any Day in 7-day Follow-up | 1871.8 (858.64)

81. Primary Outcome: Stage 1: Change From Baseline in Hematology Parameter - Leukocyte Levels
Description: Hematology parameters included hemoglobin, hematocrit, platelets, erythrocytes, neutrophils, basophils, eosinophils, monocytes, lymphocytes, leukocytes, erythrocytes mean corpuscular volume, and mean cell hemoglobin. CFB in leukocyte levels is reported in this outcome measure. Baseline is defined as the pre-infusion value in each period/stage.
Time Frame: as for outcome 21
Population: as for outcome 59
Measure: Mean (Standard Deviation); unit: 10^3 cells/μL
Arm/Group | Stage 1: SAGE-547 | Stage 1: Placebo
Number analyzed (Participants) | 25 | 25
10^3 cells/μL
  Pre-infusion | 6.976 (1.9550) | 6.972 (2.1314)
  CFB at 12-hours Follow-up: number analyzed (Participants) | 25 | 24
  CFB at 12-hours Follow-up | -0.12 (1.090) | -0.43 (0.927)

82. Primary Outcome: Stage 2: Absolute Values of Hematology Parameter - Leukocyte Levels
Description: Hematology parameters included hemoglobin, hematocrit, platelets, erythrocytes, neutrophils, basophils, eosinophils, monocytes, lymphocytes, leukocytes, erythrocytes mean corpuscular volume, and mean cell hemoglobin. Absolute values for leukocyte levels are reported in this outcome measure.
Time Frame: Stage 2: Any day in Screening period (Day -7 up to Day -1) and any day in 7-day follow up
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: 10^3 cells/μL
Arm/Group | Stage 2: SAGE-547
Number analyzed (Participants) | 17
10^3 cells/μL
  Any Day in Screening Period (Day -7 up to Day -1) | 6.928 (1.7603)
  Any Day in 7-day Follow-up | 6.688 (1.5791)

83. Primary Outcome: Stage 1: Change From Baseline in Hematology Parameter - Erythrocytes Mean Corpuscular Volume Levels
Description: Hematology parameters included hemoglobin, hematocrit, platelets, erythrocytes, neutrophils, basophils, eosinophils, monocytes, lymphocytes, leukocytes, erythrocytes mean corpuscular volume, and mean cell hemoglobin. CFB in erythrocytes mean corpuscular volume levels is reported in this outcome measure. Baseline is defined as the pre-infusion value in each period/stage.
Time Frame: as for outcome 21
Population: as for outcome 59
Measure: Mean (Standard Deviation); unit: femtoliter (fL)
Arm/Group | Stage 1: SAGE-547 | Stage 1: Placebo
Number analyzed (Participants) | 25 | 25
femtoliter (fL)
  Pre-infusion | 91.71 (3.774) | 91.72 (3.780)
  CFB at 12-hours Follow-up: number analyzed (Participants) | 25 | 24
  CFB at 12-hours Follow-up | 0.30 (0.810) | -0.03 (0.833)

84. Primary Outcome: Stage 2: Absolute Values of Hematology Parameter - Erythrocytes Mean Corpuscular Volume Levels
Description: Hematology parameters included hemoglobin, hematocrit, platelets, erythrocytes, neutrophils, basophils, eosinophils, monocytes, lymphocytes, leukocytes, erythrocytes mean corpuscular volume, and mean cell hemoglobin. Absolute values for erythrocytes mean corpuscular volume levels are reported in this outcome measure.
Time Frame: Stage 2: Any day in Screening period (Day -7 up to Day -1) and any day in 7-day follow up
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: fL
Arm/Group | Stage 2: SAGE-547
Number analyzed (Participants) | 17
fL
  Any Day in Screening Period (Day -7 up to Day -1) | 91.59 (5.264)
  Any Day in 7-day Follow-up | 91.43 (4.718)

85. Primary Outcome: Stage 1: Change From Baseline in Hematology Parameter - Mean Cell Hemoglobin Levels
Description: Hematology parameters included hemoglobin, hematocrit, platelets, erythrocytes, neutrophils, basophils, eosinophils, monocytes, lymphocytes, leukocytes, erythrocytes mean corpuscular volume, and mean cell hemoglobin. CFB in mean cell hemoglobin levels is reported in this outcome measure. Baseline is defined as the pre-infusion value in each period/stage.
Time Frame: as for outcome 21
Population: as for outcome 41
Measure: Mean (Standard Deviation); unit: picograms (pg)
Arm/Group | Stage 1: SAGE-547 | Stage 1: Placebo
Number analyzed (Participants) | 13 | 13
picograms (pg)
  Pre-infusion | 30.58 (1.540) | 30.90 (1.760)
  CFB at 12-hours Follow-up: number analyzed (Participants) | 13 | 12
  CFB at 12-hours Follow-up | 0.18 (0.468) | -0.30 (0.792)

86. Primary Outcome: Stage 2: Absolute Values of Hematology Parameter - Mean Cell Hemoglobin
Description: Hematology parameters included hemoglobin, hematocrit, platelets, erythrocytes, neutrophils, basophils, eosinophils, monocytes, lymphocytes, leukocytes, erythrocytes mean corpuscular volume, and mean cell hemoglobin. Absolute values for mean cell hemoglobin levels are reported in this outcome measure.
Time Frame: Stage 2: Any day in Screening period (Day -7 up to Day -1) and any day in 7-day follow up
Population: as for outcome 74
Measure: Mean (Standard Deviation); unit: pg
Arm/Group | Stage 2: SAGE-547
Number analyzed (Participants) | 6
pg
  Any Day in Screening Period (Day -7 up to Day -1) | 29.93 (2.890)
  Any Day in 7-day Follow-up | 29.97 (2.809)

87. Primary Outcome: Stage 1: Change From Baseline in Electrocardiogram (ECG) Parameter - QT Interval
Description: ECG parameters included QT interval, PR interval, QRS duration, QTcB interval, QTcF interval, and heart rate. CFB in QT interval is reported in this outcome measure. Baseline is defined as the pre-infusion value in each period/stage.
Time Frame: Day 1 of Stage 1 (Treatment Period 1) or on Day 10 of Stage 1 (Treatment Period 2): Pre-infusion (Baseline) and 4, 8,12 hours during infusion
Population: as for baseline characteristics
Measure: Median (Full Range); unit: milliseconds (msec)
Arm/Group | Stage 1: SAGE-547 | Stage 1: Placebo
Number analyzed (Participants) | 25 | 25
milliseconds (msec)
  Pre-infusion | 392.0 [362 to 493] | 394.0 [359 to 462]
  CFB at 4 Hours | 3.0 [-88 to 28] | -2.0 [-31 to 26]
  CFB at 8 Hours | -8.0 [-92 to 18] | -10.0 [-64 to 38]
  CFB at 12 Hours | -12.0 [-90 to 24] | -14.0 [-48 to 32]

88. Primary Outcome: Stage 2: Change From Baseline in ECG Parameter - QT Interval
Description: as for outcome 87
Time Frame: Stage 2 Day 1: Pre-infusion (Baseline) and 10 hours post-infusion
Population: as for outcome 6
Measure: Median (Full Range); unit: msec
Arm/Group | Stage 2: SAGE-547
Number analyzed (Participants) | 17
msec
  Pre-infusion: number analyzed (Participants) | 7
  Pre-infusion | 376.0 [368 to 422]
  CFB at 10 Hours: number analyzed (Participants) | 16
  CFB at 10 Hours | -1.0 [-33 to 28]

89. Primary Outcome: Stage 1: Change From Baseline in ECG Parameter - PR Interval
Description: ECG parameters included QT interval, PR interval, QRS duration, QTcB interval, QTcF interval, and heart rate. CFB in PR interval is reported in this outcome measure. Baseline is defined as the pre-infusion value in each period/stage.
Time Frame: as for outcome 87
Population: as for baseline characteristics
Measure: Median (Full Range); unit: msec
Arm/Group | Stage 1: SAGE-547 | Stage 1: Placebo
Number analyzed (Participants) | 25 | 25
msec
  Pre-infusion | 168.0 [108 to 214] | 170.0 [116 to 262]
  CFB at 4 Hours | 0.0 [-168 to 46] | -4.0 [-46 to 28]
  CFB at 8 Hours | -3.0 [-18 to 54] | -2.0 [-30 to 18]
  CFB at 12 Hours | -4.0 [-158 to 74] | -6.0 [-52 to 39]

90. Primary Outcome: Stage 2: Change From Baseline in ECG Parameter - PR Interval
Description: as for outcome 89
Time Frame: Stage 2 Day 1: Pre-infusion (Baseline) and 10 hours post-infusion
Population: as for outcome 6
Measure: Median (Full Range); unit: msec
Arm/Group | Stage 2: SAGE-547
Number analyzed (Participants) | 17
msec
  Pre-infusion: number analyzed (Participants) | 7
  Pre-infusion | 144.0 [136 to 174]
  CFB at 10 Hours: number analyzed (Participants) | 16
  CFB at 10 Hours | 2.5 [-6 to 43]

91. Primary Outcome: Stage 1: Change From Baseline in ECG Parameter - QRS Duration
Description: ECG parameters included QT interval, PR interval, QRS duration, QTcB interval, QTcF interval, and heart rate. CFB in QRS duration is reported in this outcome measure. Baseline is defined as the pre-infusion value in each period/stage.
Time Frame: Day 1 of Stage 1 (Treatment Period 1) or on Day 10 of Stage 1 (Treatment Period 2): Pre-infusion (Baseline) and 4, 8, 12 hours during infusion
Population: as for baseline characteristics
Measure: Median (Full Range); unit: msec
Arm/Group | Stage 1: SAGE-547 | Stage 1: Placebo
Number analyzed (Participants) | 25 | 25
msec
  Pre-infusion | 86.0 [72 to 236] | 85.0 [72 to 122]
  CFB at 4 Hours | 0.0 [-162 to 15] | 0.0 [-10 to 6]
  CFB at 8 Hours | 0.0 [-166 to 9] | 0.0 [-8 to 13]
  CFB at 12 Hours | 0.0 [-162 to 22] | 0.0 [-13 to 15]

92. Primary Outcome: Stage 2: Change From Baseline in ECG Parameter - QRS Duration
Description: as for outcome 91
Time Frame: Stage 2 Day 1: Pre-infusion (Baseline) and 10 hours post-infusion
Population: as for outcome 6
Measure: Median (Full Range); unit: msec
Arm/Group | Stage 2: SAGE-547
Number analyzed (Participants) | 17
msec
  Pre-infusion: number analyzed (Participants) | 7
  Pre-infusion | 90.0 [74 to 122]
  CFB at 10 Hours: number analyzed (Participants) | 16
  CFB at 10 Hours | 0.0 [-6 to 15]

93. Primary Outcome: Stage 1: Change From Baseline in ECG Parameter - QTcB Interval
Description: ECG parameters included QT interval, PR interval, QRS duration, QTcB interval, QTcF interval, and heart rate. CFB in QTcB interval is reported in this outcome measure. Baseline is defined as the pre-infusion value in each period/stage.
Time Frame: as for outcome 91
Population: as for baseline characteristics
Measure: Median (Full Range); unit: msec
Arm/Group | Stage 1: SAGE-547 | Stage 1: Placebo
Number analyzed (Participants) | 25 | 25
msec
  Pre-infusion | 412.0 [380 to 524] | 413.0 [383 to 455]
  CFB at 4 Hours | -1.0 [-111 to 18] | 1.0 [-27 to 20]
  CFB at 8 Hours | 5.0 [-115 to 28] | 0.0 [-25 to 20]
  CFB at 12 Hours | 4.0 [-108 to 78] | -1.0 [-18 to 24]

94. Primary Outcome: Stage 2: Change From Baseline in ECG Parameter - QTcB Interval
Description: as for outcome 93
Time Frame: Stage 2 Day 1: Pre-infusion (Baseline) and 10 hours post-infusion
Population: as for outcome 6
Measure: Median (Full Range); unit: msec
Arm/Group | Stage 2: SAGE-547
Number analyzed (Participants) | 17
msec
  Pre-infusion: number analyzed (Participants) | 7
  Pre-infusion | 421.0 [391 to 446]
  CFB at 10 Hours: number analyzed (Participants) | 16
  CFB at 10 Hours | 1.5 [-22 to 25]

95. Primary Outcome: Stage 1: Change From Baseline in ECG Parameter - QTcF Interval
Description: ECG parameters included QT interval, PR interval, QRS duration, QTcB interval, QTcF interval, and heart rate. CFB in QTcF interval is reported in this outcome measure. Baseline is defined as the pre-infusion value in each period/stage.
Time Frame: as for outcome 91
Population: as for baseline characteristics
Measure: Median (Full Range); unit: msec
Arm/Group | Stage 1: SAGE-547 | Stage 1: Placebo
Number analyzed (Participants) | 25 | 25
msec
  Pre-infusion | 404.0 [380 to 502] | 404.0 [389 to 451]
  CFB at 4 Hours | 2.0 [-103 to 20] | 0.0 [-24 to 18]
  CFB at 8 Hours | 1.0 [-108 to 17] | -3.0 [-17 to 20]
  CFB at 12 Hours | 1.0 [-102 to 59] | -7.0 [-17 to 23]

96. Primary Outcome: Stage 2: Change From Baseline in ECG Parameter - QTcF Interval
Description: as for outcome 95
Time Frame: Stage 2 Day 1: Pre-infusion (Baseline) and 10 hours post-infusion
Population: as for outcome 6
Measure: Median (Full Range); unit: msec
Arm/Group | Stage 2: SAGE-547
Number analyzed (Participants) | 17
msec
  Pre-infusion: number analyzed (Participants) | 7
  Pre-infusion | 406.0 [386 to 438]
  CFB at 10 Hours: number analyzed (Participants) | 16
  CFB at 10 Hours | 2.5 [-15 to 26]

97. Primary Outcome: Stage 1: Change From Baseline in ECG Parameter - Heart Rate
Description: ECG parameters included QT interval, PR interval, QRS duration, QTcB interval, QTcF interval, and heart rate. CFB in heart rate is reported in this outcome measure. Baseline is defined as the pre-infusion value in each period/stage.
Time Frame: as for outcome 91
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | Stage 1: SAGE-547 | Stage 1: Placebo
Number analyzed (Participants) | 25 | 25
bpm
  Pre-infusion | 65.0 (9.70) | 65.0 (9.09)
  CFB at 4 Hours | -1.9 (6.36) | 0.2 (4.33)
  CFB at 8 Hours | 3.3 (6.46) | 3.0 (9.05)
  CFB at 12 Hours | 5.5 (7.35) | 4.6 (7.34)

98. Primary Outcome: Stage 2: Change From Baseline in ECG Parameter - Heart Rate
Description: as for outcome 97
Time Frame: Stage 2 Day 1: Pre-infusion (Baseline) and 10 hours post-infusion
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | Stage 2: SAGE-547
Number analyzed (Participants) | 17
bpm
  Pre-infusion: number analyzed (Participants) | 7
  Pre-infusion | 72.0 (8.27)
  CFB at 10 Hours: number analyzed (Participants) | 16
  CFB at 10 Hours | -0.4 (5.97)

99. Secondary Outcome: Stage 1: Change From Baseline in Accelerometer Total Score Response
Description: Accelerometer total score response was defined as ≥30% decrease from baseline to each time point in accelerometer total score. Accelerometer total score is sum of forward outstretched postural tremor, lateral wing-beating postural tremor, and kinetic tremor scores across both sides of the body (i.e., right and left). Accelerometer was used for transducer measurement of tremor amplitude. Participants wore wireless ring motion sensor. It measured linear acceleration and angular velocity (i.e., kinesia score). Information from motion sensor data was correlated to symptoms of tremor. Kinesia (accelerometer) scores ranged from 0 to 4 in 0.5 step increments. The total score ranges from 0 to 24, higher scores indicating more severe tremors. Negative change from baseline indicated decrease in tremor. Baseline is defined as the pre-infusion value in each period/stage.
Time Frame: Stage 1 Days 1 and 10: Pre-infusion (Baseline) and 2, 4, 6, 8, 10 and 12 hours and 12-hour follow-up post-infusion
Population: Efficacy population was defined as all participants in the safety population who completed ≥12 hours of infusion and had efficacy evaluations through the 12-hour visits in both Treatment Periods 1 and 2 of Stage 1. Number analyzed = Number of participants with data available at the specific time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stage 1: SAGE-547 | Stage 1: Placebo
Number analyzed (Participants) | 25 | 25
score on a scale
  Pre-infusion: number analyzed (Participants) | 24 | 25
  Pre-infusion | 7.13 (3.902) | 7.41 (4.137)
  CFB at 2 Hours: number analyzed (Participants) | 24 | 24
  CFB at 2 Hours | -0.96 (1.373) | -1.05 (1.563)
  CFB at 4 Hours: number analyzed (Participants) | 24 | 25
  CFB at 4 Hours | -0.83 (1.876) | -0.74 (1.833)
  CFB at 6 Hours: number analyzed (Participants) | 24 | 25
  CFB at 6 Hours | -1.25 (1.943) | -0.75 (1.186)
  CFB at 8 Hours: number analyzed (Participants) | 24 | 25
  CFB at 8 Hours | -0.93 (1.903) | -1.03 (1.447)
  CFB at 10 Hours: number analyzed (Participants) | 24 | 24
  CFB at 10 Hours | -1.24 (1.814) | -0.85 (1.713)
  CFB at 12 Hours: number analyzed (Participants) | 24 | 25
  CFB at 12 Hours | -1.39 (1.436) | -0.91 (1.284)
  CFB at 12-hour Follow-up: number analyzed (Participants) | 24 | 25
  CFB at 12-hour Follow-up | 0.05 (1.498) | -0.21 (1.927)

100. Secondary Outcome: Stage 2: Change From Baseline in Accelerometer Total Score Response
Description: Accelerometer total score response was defined as ≥30% decrease from baseline to each time point in accelerometer total score. Accelerometer total score is sum of forward outstretched postural tremor, lateral wing beating postural tremor, and kinetic tremor scores across both sides of the body (i.e., right and left). Accelerometer was used for transducer measurement of tremor amplitude. Participants wore wireless ring motion sensor. It measured linear acceleration and angular velocity (i.e., kinesia score). Information from motion sensor data was correlated to symptoms of tremor. Kinesia (accelerometer) scores ranged from 0 to 4 in 0.5 step increments. The total score ranges from 0 to 24, higher scores indicating more severe tremors. Negative change from baseline indicated decrease in tremor. Baseline is defined as the pre-infusion value in each period/stage.
Time Frame: Stage 2 Day 1: Baseline and 2, 3, 4, 6, 8, 10, 12, 14 and 24 hours
Population: Efficacy population was participants from safety population, who completed ≥12 hours of infusion and had efficacy evaluations through the 12-hour visits in both Treatment Periods 1 and 2, who received study drug in Stage 2. Number analyzed = Number of participants with data available at the specific time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stage 2: SAGE-547
Number analyzed (Participants) | 17
score on a scale
  Baseline | 6.96 (4.901)
  CFB at 2 Hours: number analyzed (Participants) | 16
  CFB at 2 Hours | -1.37 (2.202)
  CFB at 3 Hours: number analyzed (Participants) | 16
  CFB at 3 Hours | -1.25 (1.890)
  CFB at 4 Hours: number analyzed (Participants) | 16
  CFB at 4 Hours | -1.57 (2.186)
  CFB at 6 Hours: number analyzed (Participants) | 16
  CFB at 6 Hours | -1.44 (2.553)
  CFB at 8 Hours: number analyzed (Participants) | 16
  CFB at 8 Hours | -2.06 (2.942)
  CFB at 10 Hours: number analyzed (Participants) | 16
  CFB at 10 Hours | -1.16 (1.809)
  CFB at 12 Hours: number analyzed (Participants) | 16
  CFB at 12 Hours | -0.89 (1.845)
  CFB at 14 Hours: number analyzed (Participants) | 16
  CFB at 14 Hours | -0.35 (1.780)
  CFB at 24 Hours: number analyzed (Participants) | 16
  CFB at 24 Hours | 0.18 (2.033)

101. Secondary Outcome: Stage 1: Change From Baseline in The Essential Tremor Rating Scale (TETRAS) Using Performance Subscale (PS) Part 4 Upper-Limb Total Scores
Description: The TETRAS PS total score was calculated as the sum of items 4 (upper-limb), 6 (Archimedes spiral), 7 (handwriting), and 8 (dot approximation). TETRAS PS upper-limb total score was calculated as the sum of the 6 separate upper-limb maneuvers assessed by the clinician: forward-outstretched postural tremor [right], forward outstretched postural tremor [left], lateral wing-beating postural tremor [right], lateral wing-beating postural tremor [left], kinetic tremor [right], kinetic tremor [left], each on a 0 (no tremor) to 4 (maximum tremor) severity scale in 0.5-point increments. TETRAS Part 4 score for both upper limbs ranged from 0 to 24, higher scores indicated more severe tremor. A negative change from baseline indicated less tremor. Baseline is defined as the pre-infusion value in each period/stage.
Time Frame: Stage 1 Days 1 and 10: Pre-infusion (Baseline) and 2, 4, 6, 8, 10 and 12 hours and 12-hour follow-up post-infusion
Population: Efficacy population was defined as all participants in the safety population who completed ≥12 hours of infusion and had efficacy evaluations through the 12-hour visits in both Treatment Periods 1 and 2 of Stage 1.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stage 1: SAGE-547 | Stage 1: Placebo
Number analyzed (Participants) | 25 | 25
score on a scale
  Pre-infusion | 9.48 (3.917) | 9.72 (3.199)
  CFB at 2 Hours | -2.10 (2.309) | -2.10 (1.860)
  CFB at 4 Hours | -2.06 (2.205) | -2.72 (2.107)
  CFB at 6 Hours | -2.94 (2.007) | -1.84 (1.553)
  CFB at 8 Hours | -2.94 (2.682) | -2.74 (1.943)
  CFB at 10 Hours | -2.94 (2.505) | -2.60 (1.898)
  CFB at 12 Hours | -3.48 (2.632) | -2.46 (2.031)
  CFB at 12-hour Follow-up | -1.38 (1.943) | -1.70 (1.507)

102. Secondary Outcome: Stage 2: Change From Baseline in TETRAS Using PS Part 4 Upper-Limb Total Scores
Description: The TETRAS PS total score was calculated as the sum of items 4 (upper-limb), 6 (Archimedes spiral), 7 (handwriting), and 8 (dot approximation). TETRAS PS upper-limb total score was calculated as the sum of the 6 separate upper-limb maneuvers assessed by the clinician: forward-outstretched postural tremor [right], forward outstretched postural tremor [left], lateral wing-beating postural tremor [right], lateral wing-beating postural tremor [left], kinetic tremor [right], kinetic tremor [left], each on a 0 (no tremor) to 4 (maximum tremor) severity scale in 0.5-point increments. TETRAS Part 4 score for both upper limbs ranged from 0 to 24, higher scores indicated more severe tremor. A negative change from baseline indicated less tremor.
Time Frame: Stage 2 Day 1: Baseline and at 2, 3, 4, 6, 8, 10, 12, 14 and 24 hours
Population: as for outcome 100
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stage 2: SAGE-547
Number analyzed (Participants) | 17
score on a scale
  Baseline | 9.24 (1.977)
  CFB at 2 Hours: number analyzed (Participants) | 16
  CFB at 2 Hours | -1.66 (2.173)
  CFB at 3 Hours: number analyzed (Participants) | 16
  CFB at 3 Hours | -2.44 (2.542)
  CFB at 4 Hours: number analyzed (Participants) | 16
  CFB at 4 Hours | -3.25 (2.550)
  CFB at 6 Hours: number analyzed (Participants) | 16
  CFB at 6 Hours | -2.66 (2.612)
  CFB at 8 Hours: number analyzed (Participants) | 16
  CFB at 8 Hours | -3.16 (2.809)
  CFB at 10 Hours: number analyzed (Participants) | 16
  CFB at 10 Hours | -2.19 (1.642)
  CFB at 12 Hours: number analyzed (Participants) | 16
  CFB at 12 Hours | -1.25 (1.602)
  CFB at 14 Hours: number analyzed (Participants) | 16
  CFB at 14 Hours | -0.66 (1.091)
  CFB at 24 Hours: number analyzed (Participants) | 16
  CFB at 24 Hours | -0.84 (1.850)

103. Secondary Outcome: Stage 1: Change From Baseline in Stanford Sleepiness Scale (SSS) Score
Description: SSS is a participant-rated scale designed to quickly assess how alert a participant was feeling. Degrees of sleepiness and alertness were rated on a scale of 1 to 7, where the lowest score of '1' indicated the participant was 'feeling active, vital, alert, or wide awake' and the highest score of '7' indicated the participant was 'no longer fighting sleep, sleep onset soon; having dream-like thoughts'. Baseline is defined as the pre-infusion value in each period. A negative change from baseline indicated less sleepiness.
Time Frame: Stage 1 Day 1 and 10: Pre-infusion (Baseline) and 2, 4, 6, 8, 10 and 12 hours and 12-hour follow-up post-infusion
Population: Efficacy population was defined as all participants in the safety population who completed ≥12 hours of infusion and had efficacy evaluations through the 12-hour visits in both Treatment Periods 1 and 2 of Stage 1. Overall number of participants analyzed = Number of participants analyzed in this outcome measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stage 1: SAGE-547 | Stage 1: Placebo
Number analyzed (Participants) | 24 | 25
score on a scale
  Pre-infusion | 1.6 (0.77) | 1.6 (0.76)
  CFB at 2 Hours | 0.3 (1.37) | 0.0 (0.41)
  CFB at 4 Hours | 0.3 (1.40) | 0.1 (0.53)
  CFB at 6 Hours | 0.7 (1.09) | 0.1 (0.83)
  CFB at 8 Hours | 0.1 (1.08) | 0.0 (0.82)
  CFB at 10 Hours | 0.3 (1.40) | 0.2 (0.93)
  CFB at 12 Hours | 0.2 (0.87) | -0.0 (0.89)
  CFB at 12-hour Follow-up | -0.1 (0.54) | -0.2 (0.75)

104. Secondary Outcome: Stage 2: Change From Baseline in Stanford Sleepiness Scale (SSS) Score
Description: as for outcome 103
Time Frame: Stage 2 Day 1: Baseline and at 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 14 and 24 hours
Population: Efficacy population was participants from safety population who completed ≥12 hours of infusion and had efficacy evaluations through the 12-hour visits in both Treatment Periods 1 and 2, who received study drug in Stage 2. Number analyzed = Number of participants with data available at the specific time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stage 2: SAGE-547
Number analyzed (Participants) | 17
score on a scale
  Baseline | 1.5 (0.62)
  CFB at 1 Hour | 0.4 (1.12)
  CFB at 2 Hours: number analyzed (Participants) | 16
  CFB at 2 Hours | 1.4 (1.09)
  CFB at 3 Hours: number analyzed (Participants) | 16
  CFB at 3 Hours | 2.5 (2.10)
  CFB at 4 Hours: number analyzed (Participants) | 16
  CFB at 4 Hours | 3.1 (1.81)
  CFB at 5 Hours: number analyzed (Participants) | 16
  CFB at 5 Hours | 3.3 (2.02)
  CFB at 6 Hours: number analyzed (Participants) | 16
  CFB at 6 Hours | 3.3 (1.91)
  CFB at 7 Hours: number analyzed (Participants) | 16
  CFB at 7 Hours | 2.6 (1.79)
  CFB at 8 Hours: number analyzed (Participants) | 16
  CFB at 8 Hours | 2.4 (1.86)
  CFB at 9 Hours: number analyzed (Participants) | 16
  CFB at 9 Hours | 2.3 (1.91)
  CFB at 10 Hours: number analyzed (Participants) | 16
  CFB at 10 Hours | 2.0 (1.97)
  CFB at 11 Hours: number analyzed (Participants) | 16
  CFB at 11 Hours | 0.1 (0.85)
  CFB at 12 Hours: number analyzed (Participants) | 16
  CFB at 12 Hours | -0.3 (0.86)
  CFB at 14 Hours: number analyzed (Participants) | 16
  CFB at 14 Hours | 0.3 (1.44)
  CFB at 24 Hours: number analyzed (Participants) | 16
  CFB at 24 Hours | -0.3 (0.86)

105. Secondary Outcome: Stage 1: Maximum Peak Plasma Concentration (Cmax) of SAGE-547
Time Frame: Stage 1: Pre-infusion and after the start of infusion at 30 and 40 minutes and at 1, 1.5, 2, 4, 6, 8, 10, 12, 12.5, 12.75, 13, 13.5, 14, 16 and 24 hours
Population: Pharmacokinetic (PK) population was defined as all safety population participants who completed at least 12 hours of SAGE-547 infusion in Treatment Period 1 or Treatment Period 2 of Stage 1 with sufficient plasma concentrations for PK evaluation.
Measure: Mean (Standard Deviation); unit: nanograms per milliliter (ng/mL)
Arm/Group | Stage 1: SAGE-547
Number analyzed (Participants) | 25
nanograms per milliliter (ng/mL) | 84.3 (28.2)

106. Secondary Outcome: Stage 2: Maximum Peak Plasma Concentration (Cmax) of SAGE-547
Time Frame: Stage 2: Pre-infusion and at 30, 60, 90 and 120 minutes and at 2.5, 3, 4, 5, 6, 7, 8, 9, 10, 10.5, 10.75, 11, 11.5, 12, 14, 16 and 24 hours after start of the infusion
Population: PK population was participants from safety population, who completed at least 12 hours of SAGE-547 infusion in Treatment Period 1 or Treatment Period 2 with sufficient plasma concentrations for PK evaluation, who received study drug in Stage 2.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Stage 2: SAGE-547
Number analyzed (Participants) | 17
ng/mL | 152 (36)

107. Secondary Outcome: Stage 1: Time to Maximum Peak Plasma Concentration (Cmax) of SAGE-547
Time Frame: as for outcome 105
Population: PK population was defined as all safety population participants who completed at least 12 hours of SAGE-547 infusion in Treatment Period 1 or Treatment Period 2 of Stage 1 with sufficient plasma concentrations for PK evaluation.
Measure: Median (Full Range); unit: hours
Arm/Group | Stage 1: SAGE-547
Number analyzed (Participants) | 25
hours | 10 [1 to 12.483]

108. Secondary Outcome: Stage 2: Time to Maximum Peak Plasma Concentration (Cmax) of SAGE-547
Time Frame: as for outcome 106
Population: as for outcome 106
Measure: Median (Full Range); unit: hours
Arm/Group | Stage 2: SAGE-547
Number analyzed (Participants) | 17
hours | 6 [2.967 to 9.05]

109. Secondary Outcome: Stage 1: Area Under the Plasma Concentration Time Curve up to the Time of the Last Quantifiable Sample (AUClast) of SAGE-547
Time Frame: as for outcome 105
Population: as for outcome 107
Measure: Mean (Standard Deviation); unit: nanograms*hours per milliliter (ng*h/mL)
Arm/Group | Stage 1: SAGE-547
Number analyzed (Participants) | 25
nanograms*hours per milliliter (ng*h/mL) | 654 (251)

110. Secondary Outcome: Stage 2: Area Under the Plasma Concentration Time Curve up to the Time of the Last Quantifiable Sample (AUClast) of SAGE-547
Time Frame: Day 1: Pre-infusion and at 30, 60, 90 and 120 minutes and at 2.5, 3, 4, 5, 6, 7, 8, 9, 10, 10.5, 10.75, 11, 11.5, 12, 14, 16 and 24 hours after start of the infusion
Population: as for outcome 106
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Stage 2: SAGE-547
Number analyzed (Participants) | 17
ng*h/mL | 1310 (300)

111. Secondary Outcome: Stage 1: Area Under the Concentration-Time Curve From Time 0 to Infinity (AUC0-inf) of SAGE-547
Time Frame: as for outcome 105
Population: as for outcome 107
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Stage 1: SAGE-547
Number analyzed (Participants) | 25
ng*h/mL | 716 (286)

112. Secondary Outcome: Stage 2: Area Under the Concentration-Time Curve From Time 0 to Infinity (AUC0-inf) of SAGE-547
Time Frame: as for outcome 106
Population: as for outcome 106
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Stage 2: SAGE-547
Number analyzed (Participants) | 17
ng*h/mL | 1380 (300)

113. Secondary Outcome: Stage 1: Clearance (CL) of SAGE-547
Description: Clearance is defined as the volume of plasma from which a substance is completely removed per unit time.
Time Frame: as for outcome 105
Population: as for outcome 107
Measure: Mean (Standard Deviation); unit: liters per hour per kilogram (L/h/kg)
Arm/Group | Stage 1: SAGE-547
Number analyzed (Participants) | 25
liters per hour per kilogram (L/h/kg) | 1.09 (0.41)

114. Secondary Outcome: Stage 2: Clearance (CL) of SAGE-547
Description: Clearance is defined as the volume of plasma from which a substance is completely removed per unit time.
Time Frame: as for outcome 106
Population: as for outcome 106
Measure: Mean (Standard Deviation); unit: L/h/kg
Arm/Group | Stage 2: SAGE-547
Number analyzed (Participants) | 17
L/h/kg | 1.07 (0.28)

115. Secondary Outcome: Stage 1: Terminal Half-Life (t½) of SAGE-547
Description: Terminal half-life is defined as the time required to divide the plasma concentration by two after reaching pseudo-equilibrium.
Time Frame: as for outcome 105
Population: as for outcome 107
Measure: Median (Full Range); unit: hours
Arm/Group | Stage 1: SAGE-547
Number analyzed (Participants) | 25
hours | 5.6 [1.8 to 12.8]

116. Secondary Outcome: Stage 2: Terminal Half-Life (t½) of SAGE-547
Description: as for outcome 115
Time Frame: as for outcome 106
Population: as for outcome 107
Measure: Median (Full Range); unit: hours
Arm/Group | Stage 2: SAGE-547
Number analyzed (Participants) | 17
hours | 7.6 [4.8 to 9.5]

ADVERSE EVENTS:
Time Frame: Stage 1: Up to 30 days after last infusion (up to Day 40); Stage 2: Up to 30 days after last infusion (up to Day 31)
Description: Safety population for Stage 1 included all participants admitted into the inpatient unit who met all eligibility criteria, signed an informed consent, and who began infusion with SAGE-547 or placebo in Treatment Period 1 of Stage 1. The safety population for Stage 2 included all participants admitted into the inpatient unit who met all eligibility criteria, signed an informed consent, and who began infusion with SAGE-547 or placebo in Treatment Period 1, who received study drug in Stage 2.
Arm/Group | Stage 1: SAGE-547 | Stage 1: Placebo | Stage 2: SAGE-547
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/25 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25 | 0/17
Other Adverse Events (participants affected / at risk) | 1/25 | 3/25 | 8/17
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Stage 1: SAGE-547 (N=25) | Stage 1: Placebo (N=25) | Stage 2: SAGE-547 (N=17)
Fatigue (General disorders) | 1 | 0 | 4
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 2 | 3
Headache (Nervous system disorders) | 0 | 1 | 1
Sedation (Nervous system disorders) | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI can either be a party and subject to the same restrictions as the institution, or if not a party, the restrictions are described on the face of the contract (i.e., PI is a contractor of the institution; PI is part of a larger group of study personnel; institution has contracted with or otherwise bound all study personnel under confidentiality obligations and requirements to vest intellectual property to the institution).